

Valeant Pharmaceuticals North America

VRX-RET-E22-304

A multicenter, open-label, long-term, safety, tolerability and efficacy study of retigabine in adult epilepsy patients with partial-onset seizures (Extension of Study VRX-RET-E22-302)

Statistical Analysis Plan

Version 2.0 [Final] Date: February 26, 2007

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America VRX-RET-E22-304

Statistical Analysis Plan Version 2.0 [Final]

#### SIGNATURE PAGE

Prepared by:

26 FEB 2008 Date

Director, B&P

PAREXEL International

Reviewed and Approved by:

PhD

February 26, 2008
Date

Director, Biostatistics

Valeant Pharmaceuticals North America

26 - Feb - 2008 Date

Director, Clinical Operations

Valeant Pharmaceuticals North America

Feb 26, 2008

MD

Sr. VP, Global Drug Development Valeant Pharmaceuticals North America

MD, PhD

VP, Global Safety and Pharmacovigilance Valeant Pharmaceuticals North America 26 Feb 2008 Date

101

BSc, PhD, PMP

VP, Global Regulatory Sciences Valeant Pharmaceuticals North America 26 Feb 2008

Date

MD, PhD, ScM

Chief Medical Officer & VP, Global Medical Affairs Valeant Pharmaceuticals North America 26 Feb 2008 "

Date

# **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 5 |
|---|---|---|
| 2 | STUDY OBJECTIVES | 6 |
| 3 | INVESTIGATIONAL PLAN | |
| | 3.1 Overall Study Design and Plan | |
| | 3.2 Efficacy and Safety Variables | |
| | 3.2.1 Efficacy Assessments. | |
| | 3.2.2 Safety Assessments | |
| | 3.2.3 Quality of Life Assessments | |
| 4 | STATISTICAL METHODS | |
| | 4.1 Study Patients | |
| | 4.1.1 Disposition of Patients | |
| | 4.1.2 Analysis Populations. | |
| | 4.2 Demographic and Other Baseline Characteristics | |
| | 4.3 General Considerations | |
| | 4.4 Efficacy Evaluation | |
| | 4.5 Safety Evaluation | |
| | 4.5.1 Extent of Exposure | |
| | 4.5.2 Adverse Events | |
| | 4.5.3 Deaths, Serious Adverse Events, and Other Significant Adverse Events. | |
| | 4.5.4 Clinical Laboratory Evaluation | |
| | 4.5.5 Vital Signs, Physical Findings and Other Observations Related to Safety | |
| | 4.5.5.1 Vital Sign Measurements | |
| | 4.5.5.2 ECG | |
| | 4.5.5.3 Physical and Neurological Examination | |
| | 4.5.5.4 AUA Symptom Index | |
| | 4.5.5.5 Post-void Residual (PVR) Bladder Ultrasound | |
| | 4.5.6 Concomitant Medications | |
| | 4.6 Quality of Life in Epilepsy (QOLIE-31-P) | 21 |
| | 4.7 Determination of Sample Size | |
| | 4.8 Changes in the Conduct of the Study or Planned Analysis | 21 |
| 5 | REFERENCES | |
| 6 | REPORTING OUTPUT | 21 |
| 7 | LIST OF TABLES | |
| 8 | LIST OF FIGURES | 27 |
| 9 | LIST OF PATIENT DATA LISTINGS | 28 |
| 10 | TABLE SHELLS | |
| 11 | FIGURE SHELLS | |
| 12 | PATIENT DATA LISTING SHELLS | 89 |

# LIST OF ABBREVIATIONS

| AE | Adverse event |
|-------------------------------|----------------------------------------------|
| AED | Antiepileptic drug |
| ALT | Alanine transaminase (SGPT) |
| AST | Aspartate transaminase (SGOT) |
| AUA | American Urological Association |
| BMI | Body mass index |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| CRA | Clinical monitor |
| CRF | Case Report Form |
| ECG | Electrocardiogram |
| ICH | International Conference of Harmonization |
| MedDRA® | Medical Dictionary for Regulatory Activities |
| ODS | Output Delivery System |
| OLE | Open-label extension |
| PVR | Post-void Residual |
| QTc | QT correction |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| $\mathrm{SAS}^{^{\circledR}}$ | Statistical Analysis Software |
| SD | Standard deviation |
| TEAE | Treatment-emergent adverse event |
| TID | Three time a day |
| WBC | White blood cell |
| WHO | World Health Organization |

#### 1 INTRODUCTION

Epilepsy is among the most common neurological disorders, affecting approximately 50 million people worldwide. Classical antiepileptic drugs (AEDs) currently provide satisfactory seizure control in approximately 70% of patients; however, the remaining 30% of epilepsy patients are refractory to treatment. The partial onset seizure is the most common type of seizure that is uncontrolled in adult patients. The introduction of new (e.g., vigabatrin. lamotrigine, gabapentin. topiramate. oxcarbazepine, zonisamide, and felbamate) during the last decade has increased therapeutic possibilities. However, data from recent clinical trials demonstrate that none of the newer AEDs provides adequate seizure control in all patients. The treatment of patients that do not respond to current AEDs remains a problem and motivates the continued search for compounds with high antiepileptic potential and low rates of side effects.

Retigabine (GKE-841 or D-23129), N-[2-amino-4(4-fluorobenzylamino)-phenyl] carbamic acid ethyl ester, is a new chemical entity discovered by ASTA Medica, Germany, and was acquired by Valeant Research & Development (Valeant) for development as an AED for the treatment of partial onset seizures. It is a deaza analog of flupirtine, currently marketed in some regions as a centrally acting analgesic with ancillary muscle relaxing properties.

Two Phase 3 studies (VRX-RET-E22-301 and VRX-RET-E22-302) to compare the efficacy and safety of retigabine (600 mg/day, 900 mg/day, or 1200 mg/day) to placebo as an adjunctive therapy in refractory patients with partial-onset seizures are currently being conducted. These studies are randomized, double-blind, placebo-controlled, multicenter, parallel-group trials enrolling a total of approximately 790 patients, globally. Because of the serious nature of epilepsy, the retigabine clinical program had foreseen that all patients who enter and complete a Phase 3 study with retigabine will be given the opportunity to continue treatment, if they consent and if the Principal Investigator feels they can benefit from continued retigabine treatment. Hence, an open-label extension protocol was designed for each double-blind study.

This study is the open-label extension of the Phase 3 Study VRX-RET-E22-302. VRX-RETE22-302 is a randomized, double-blind, placebo-controlled, parallel-group, multicenter, study of 900 mg/day and 600mg/day retigabine versus placebo. During the 4-week titration phase patients are titrated to the target dose. 510 patients are expected to be randomized to treatment. A 12-week maintenance phase follows. All patients who wish to enter the open-label extension protocol will enter a 4-week transition phase in which their dose will be titrated to 300 mg TID in order to maintain the blind to the maximum extent. Thereafter, the patients could enter this extension study (Study VRX-RET-E22-304). Patients who do not wish to enter the open-label extension protocol will have their dose tapered over a 3-week period.

This Statistical Analysis Plan (SAP) was created according to Protocol VRX-RET-E22-304, Amendment 1 (July 2, 2007).

Filename: 87272 304 SAP v2 final

#### 2 STUDY OBJECTIVES

# Primary Objective

To evaluate the safety and tolerability of long-term therapy with retigabine administered as adjunctive therapy in adult epilepsy patients with partial-onset seizures, who completed the double-blind Study VRX-RET-E22-302.

# Secondary Objective

To evaluate efficacy of long-term treatment with retigabine and patient quality of life, evaluated through the QOLIE-31-P questionnaire.

#### 3 INVESTIGATIONAL PLAN

### 3.1 Overall Study Design and Plan

This is an open-label extension study of the placebo controlled, double-blind Study VRXRET-E22-302. Patients will be treated with 600 - 1200 mg/day of retigabine as an adjunct therapy to their current antiepileptic medications (AEDs) or vagal nerve stimulation as established in Study VRX-RET-E22-302. Following completion of the Transition Phase of the double-blind study (Study VRX-RET-E22-302), treatment in this open-label extension study will be continued until retigabine is approved and commercially available, or until the program is discontinued, followed by a 3-week tapering period and a 30 day post-study period for collection of adverse events.

# 3.2 Efficacy and Safety Variables

A study flow chart summarizing all study procedures can be found in Table 1.

#### 3.2.1 Efficacy Assessments

Patients will keep a seizure diary throughout the study. The anticonvulsant efficacy of retigabine will be evaluated by comparison of baseline seizure frequency (obtained during the 8-week baseline period of Study VRX-RET-E22-302) with seizure frequency obtained during retigabine therapy in this open-label extension study (VRX-RET-E22-304). The primary efficacy variable is the percentage change in the monthly seizure rate from the baseline phase to the open-label treatment phase. The proportion of responders (patients experiencing  $\geq$  50% reduction in seizure frequency) from baseline to the open-label treatment phase will be evaluated.

**Table 1: Study Flow Chart** 

| | Baseline <sup>1</sup> | | C | Open-l | _abel E | Extens | ion-Fir | st Yea | ar <sup>2,3</sup> | | O | oen-La | bel Ex | tensio | n-Sec | ond |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedures | | | | | | | | | | | | | ar arra | | | |
| Visit | 0 | 1 | 1a <sup>9</sup> | 2 | 2a <sup>9</sup> | 3 | 3a <sup>9</sup> | 4 | 4a <sup>9</sup> | 5 <sup>4</sup> | 6 | 7 | 8 <sup>4</sup> | 9 | 10 | 11 <sup>4</sup> |
| Month in Study | 0 | 1 | 2 | 3 | 4 | 6 | 8 | 9 | 10 | 12 | 16 | 20 | 24 | 28 | 32 | 36 |
| Eligibility /ICF | Χ | | | | | | | | | | | | | | | |
| Physical & Neuro Exam | Χ | | | | | | | | | Χ | | | Х | | | Χ |
| Brief Neuro Exam | | Χ | | Χ | | Χ | | Χ | | | Χ | Х | | Х | Х | |
| Vital Signs (BP,HR,&Temp)<br>&Wt <sup>5</sup> | X | Х | | Х | | х | | х | | Х | Х | х | Х | Х | Х | Х |
| 12 Lead ECG | Χ | Х | | Х | | Х | | Х | | Х | | | Х | | | Х |
| Blood Chem and Hematology | Х | Х | | Х | | Х | | Х | | Χ | Х | Х | Х | Х | Х | Х |
| Hematological Evaluation | | | Χ | | Χ | | Χ | | Χ | | | | | | | |
| Urinalysis (including Microscopy) | Х | Х | | X | | X | | x | | Х | Х | x | х | Х | Х | х |
| AUA Symptom Index <sup>7</sup> | Х | Х | | Х | | | | | | Χ | | | | | | |
| PVR Bladder Ultrasound | Χ | Х | | Χ | | | | | | Χ | | | | | | |
| Serum Preg Test <sup>6</sup> | Х | | | | | | | | | Χ | | | Χ | | | Χ |
| Urine Preg Test <sup>6</sup> | Х | | | | | | | | | | | | | | | |
| Seizure Diary Review | Χ | Χ | | Χ | | Х | | Х | | Χ | Χ | Х | Х | Х | Х | Х |
| AE Evaluation | Χ | Х | | Χ | | Х | | Х | | Χ | Χ | Х | Х | Х | Х | Х |
| Concomitant Medication | Χ | Χ | | Χ | | Х | | Х | | Χ | Χ | Х | Х | Х | Х | Х |
| QOLIE-31-P Qx | Χ | | | Χ | | Χ | | Χ | | Χ | | | Х | | | Χ |
| Dispense OLE Study Meds <sup>8</sup> | Χ | Х | | Χ | | Х | | Χ | | Χ | Х | Х | Х | Х | Х | Χ |
| Collected Returned OLE Study Meds | | Х | | Х | | Х | | Х | | Х | Х | Х | Х | Х | Х | Х |

Filename: 87272\_304\_SAP\_v2\_final

 $\infty$ 

# 9


## **Table 1: Study Flow Chart (continued)**

- 1. Baseline for the open-label extension study corresponds to the assessments performed at the last visit of the Maintenance phase (Visit 9) of Study VRX-RET-E22-302 for all patients. The final, baseline eligibility assessment for the open-label extension study, including obtaining informed consent and dispensing open-label study medication will be performed at the last visit of the Transition phase (Visit 11) of Study VRX-RET-E22-302.
- 2. Study Visit 1 will have a window range of ±3 days. After Study Visit 1, all remaining study visits will have a window range of 7 days around that visit day to accommodate individual schedules. Each study month will be defined as 30 calendar days. If a patient visit occurs outside the visit window, the study clinical monitor (CRA) should be notified and the reason for the deviation noted. An attempt should be made to ensure that the patient returns for subsequent visits on schedule using the last visit of the Transition phase (Visit 11) of Study VRX-RET-E22-302, which corresponds to the final, Baseline eligibility visit for the open-label extension study.
- 3. This open-label extension study will be continued until retigabine is approved and commercially available, or until the program s discontinued, followed by a 3-week tapering period and a 30 day post-study period for collection of adverse events. After the first year, the study visits will occur every 4 months (3 visits per year). After the first year, the assessments for the first 2 study visits of each year (e.g. Visits 6, 7, 9 and 10) will be identical, and the assessments for the last study visit of each year (e.g. Visits 8 and 11) will be identical.
- 4. All patients who discontinue early from study treatment during the open-label extension study will have their study medication tapered over a 3-week period, reducing their daily dose by one third per week, and then return for a final visit. Patients who discontinue early during the first year of the open-label extension study will complete all assessments and evaluations scheduled for Study Visit 5. Patients who discontinue early during the second year of the open-label extension study will complete all assessments and evaluations scheduled for Study Visit 8. Patients who discontinue early during the third year of the open-label extension study will complete all assessments and evaluations scheduled for Study Visit 11. Also, all adverse events should be followed and collected up to until 30 days after administration of the last dose of study drug (end of study drug taper-off).
- 5. Supine and standing blood pressure, heart rate.
- 6. In addition to the scheduled pregnancy tests, a pregnancy test should be performed during the study whenever a woman's menstrual period is 5 days late.
- 7. The AUA Symptom Index and the PVR bladder ultrasound will only be performed during the first year of the open-label extension study (Visits 1, 2, and 5).
- 8. Dispensation of study medication is not applicable at the final study visit, if a patient has discontinued early or completed the open-label extension study.
- 9. Study visits added per FDA comments that the open label extension trial should include more frequent hematological monitoring. These are now in-line with the hematological monitoring frequencies per the VRX-RET-E22-302, double-blind trial.

## 3.2.2 Safety Assessments

Safety assessments will be evaluated, based on reports of AEs and results of vital signs (supine and standing blood pressure, pulse, and temperature), weight, clinical laboratory evaluations (blood chemistries, hematology and urinalysis including microscopy), a 12-lead ECG, and physical and neurological examinations. Post-void residual (PVR) bladder ultrasounds to assess urinary retention and the American Urological Association (AUA) Symptom Index to assess urinary voiding function will also be performed during the first year of the open-label extension study.

# 3.2.3 Quality of Life Assessments

The QOLIE-31-P (Version 2.0) will be utilized to assess quality of life. The QOLIE-31-P assessment must be completed by the patients. Patients who are cognitively impaired and cannot complete the QOLIE-31-P assessment may still participate in the study, by obtaining a waiver for QOLIE-31-P completion from the study medical monitor.

#### 4 STATISTICAL METHODS

#### 4.1 Study Patients

## 4.1.1 Disposition of Patients

Patients are free to discontinue their participation in the study at any time and without prejudice to further treatment at their local site. The Investigator must withdraw any patient from the study if that patient requests to be withdrawn. Patients withdrawn from the study will not be replaced, regardless of the reason for withdrawal. The patient's participation in this study may be discontinued due to the following reasons:

- Patient experiences an intolerable AE.
- Investigator decides patient has an "unsatisfactory response efficacy."
- Patient becomes pregnant.
- Patient is unwilling or unable to continue the study.
- Patient is non-compliant with study procedures.
- Patient needs medication not allowed in the protocol.
- Any clinically significant change in patient's medical condition.
- Persistent ALT or aspartate aminotransferase (AST) above 3 times the ULN; will be confirmed by repeating laboratory assessment within 1 week.
- ALT or AST levels are above 5 times the ULN at any time during the study.
- Confirmed QTc prolongation defined as QTc (Bazett's) >500 msec or an increase in QTc (Bazett's) of >60 msec from baseline.

- Investigator decides that withdrawal from the study is in the best interest of the patient.
- Request of the Sponsor.
- Hematological reasons or infections for all such patients, the investigator shall report these in an expedited manner, whether or not they are considered serious or unexpected.

A summary of the number and percentage of discontinuations by primary reason will be provided together with descriptive statistics for the time until treatment discontinuation (days).

A by-patient listing of patient withdrawal/study completion details will also be provided.

# 4.1.2 Analysis Populations

The Safety Population is defined as all patients who successfully completed the transition phase of Study VRX-RET-E22-302 and were enrolled into the long-term study VRX-RET-E22-304. The Transition phase is the phase of Study VRX-RET-E22-302 during which patients were adjusted to a 300 mg TID dose.

There will be no other population for this study.

## 4.2 Demographic and Other Baseline Characteristics

Demographic and baseline characteristics were not collected as part of the VRX-RET-E22-304 case report form (CRF). For the following summaries of demographic and other baseline characteristics, unless otherwise noted, the last recorded value prior to commencement of study treatment in the VRX-RET-E22-302 study will be used as baseline.

A summary of the following demographic variables will be presented at baseline:

- age
- sex
- race
- weight
- height
- body mass index (BMI)
- duration of partial and generalized seizures, separately
- type of onset of partial and generalized seizures, separately

- Baseline seizure type cohorts
- number of background AEDs
- number of patients using Vagal Nerve Stimulators
- CGI severity baseline scores

A patient's age in years will be calculated as the number of completed years between the date of the informed consent for the VRX-RET-E22-302 study and date of birth (i.e. date of informed consent minus date of birth divided by 365.25). Age, weight and BMI will be summarized using continuous descriptive statistics. The number and percentage of patients in each sex category (male and female), and each race category (Caucasian, African-American, Hispanic, Asian and Other), will be reported using categorical descriptive statistics.

Duration of partial and generalized epilepsy is defined as the difference between Year of Onset recorded in Epilepsy History and year of Visit 1 (screening) for the VRX-RET-E22-302 study. The duration of partial epilepsy will be summarized using continuous descriptive statistics.

By-patient listings of all demographic data and baseline characteristics will also be provided.

#### 4.3 General Considerations

Study day is defined as the number of days relative to Day 0 (i.e., the start of study treatment in the double-blind study VRX-RET-E22-302), computed as (the date – Day 0 date+1).

Continuous data that are assumed to be normally distributed will be summarized in terms of the mean, standard deviation (SD), median, minimum, maximum and number of observations. Continuous data that are expected to be skewed will be presented in terms of the maximum, upper quartile, median, lower quartile, minimum and number of observations. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean, SD, median, lower quartile and upper quartile will be reported to one more decimal place than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be four for any summary statistic.

Categorical data will be summarized in terms of the number of patients providing data at the relevant time point (n), frequency counts and percentages. Percentages will be presented to one decimal place. Percentages will not be presented for zero counts. Percentages will be calculated using n as the denominator.

# 4.4 Efficacy Evaluation

"Monthly total partial seizure" as well as "monthly total seizure" rates will be calculated for the entire open-label part of Study VRX-RET-E22-304 and statistically described. "Monthly total partial seizure" rate is defined as the sum of total partial seizures throughout the open-label portion (of Study VRX-RET-E22-304), divided by open-label duration in days, standardized by 28 days (1 month). "Monthly total seizure" rate is defined as the sum of partial and generalized (or unclassified) seizures throughout the open-label duration in days, standardized by 28 days (1 month).

Monthly total partial seizure rates observed during the open-label extension period will be compared to the monthly total seizure rates observed during the Baseline phase of the double-blind study VRX-RET-E22-302. The baseline monthly total seizure rates will only be derived for patients who enter this open-label extension and have a monthly total partial seizure rate during the open-label extension period. The percent change in monthly total partial seizure rates from the Baseline phase will be classified into <0, [0, 25), [25, 50), [50, 75), [75, 100] with a description of the frequencies. The responder rate during the open-label study (defined as a reduction in seizure frequency ≥50%) will also be summarized using descriptive statistics.

The monthly total partial seizure rates compared to the baseline monthly total partial seizure rate will be presented cumulatively for each timepoint (months 1, 3, 6, 9, 12, 16, 20, 24, 28, 32 and 36) during the open label extension period and separately for eleven cohorts of patients treated with retigabine for at least 1, 3, 6, 9, 12, 16, 20, 24, 28, 32 and 36 months. In each cohort, patients will be followed for entire indicated duration of treatment. For example, patients in the 36-month cohort will also be part of the shorter-duration cohorts.

A similar analysis will be repeated for the responder rate during the open-label study.

A plot of the median percent reduction from baseline in seizure frequency over time by duration of treatment will also be produced.

The number of seizure free days, in percent to the individual duration of the open-label treatment, will be calculated and summarized using descriptive statistics. "Percent seizure free days" is defined as the number of days without any seizures (partial or generalized) divided by open-label duration in days, in percent. This percentage will be classified into [0, 25), [25, 50), [50, 75), [75, 95), [95,100), [=100] and described statistically. The most upper class represents completely seizure free patients, the next class almost seizure free patients.

Additionally, the proportion of subjects who become seizure free for 6 and 12 month rolling intervals will also be determined. That is, a subject who becomes seizure free for any 6 month period of time will qualify for the 6 month metric. A subject who becomes seizure free for any 12 month period of time will qualify for both the 6 month and 12 month metric.

## 4.5 Safety Evaluation

# 4.5.1 Extent of Exposure

Exposure Daily Dose is defined as the mean value of daily dosages of study drug, that is total dosage taken by a patient divided by number of days the patient participated in the study. The total dosage is defined as sum of the recorded doses in the Study Medication and Dose Change Log for each visit. The number of days patient participated in this study is defined as the period from the first dose date (Day 0) to the last recorded dose date. Descriptive statistics of the exposure daily dose of this study will be presented.

Extent of exposure is defined as the total number of days a patient is exposed to study drug. In calculation, the extent of exposure equals the total number of days from the first dose date (Day 0) to the last recorded dose date. If a patient is lost to follow-up, but the drug accountability log confirms that the patient has taken study drug, the last visit date of the treatment period will be used for calculation of extent of exposure. For better description, extent of exposure (in weeks) will also be categorized ( $\leq 1$ , (1-3], (3-6], (6-9], (9-12], (12-16], (16-20], (20-24], (24-28], (28-32], (32-36], >36). Descriptive statistics for extent of exposure categorized by weeks will additionally be presented.

A by-patient listing of detailed exposure daily dose, dose modifications and extent of exposure to study drug will be provided. Any extreme values for both the exposure daily dose and the extent of exposure to study medications will be reported in the listings, in case that happens.

#### 4.5.2 Adverse Events

Adverse events (AEs) are monitored from the start of this extension study (informed consent provided by patient at the Baseline visit) until 30 days after administration of the last dose of study drug (end of study drug taper-off).

The AEs will be coded using the most recent Medical Dictionary for Regulatory Activities (MedDRA), Version 9.1. The number and percentage of patients experiencing at least one adverse event will be summarized overall and by body system and preferred term. In any given body system or preferred term patients will only be counted once. Adverse events will further be categorized and summarized by severity and study drug relationship. If the same event for a patient has two different severities, the worst will be taken.

Abnormal laboratory values do not themselves represent adverse events unless they:

- are indicative of a disease or defect, e.g. reduced hematocrit resulting in anemia;

- necessitate intervention, e.g., administration of packed red blood cells or other therapies; and
- result in dose reduction or permanent discontinuation of the drug product.

Worsening of seizure frequency will not be considered an AE but will be captured in the efficacy analysis. Those patients who discontinue their treatment prematurely either during the double-blind period or choose not to enter the open-label extension study should be tapered off their study treatment gradually and will be closely monitored by scheduled clinic visits for worsening of their seizure frequency during this period.

Adverse events will be graded for intensity. An intensity category of mild, moderate, or severe, is defined as

Mild Causing no limitation of usual activities; the patient may experience

slight discomfort

Moderate Causing some limitation of usual activities; the patient may experience

annoying discomfort

Severe Causing inability to carry out usual activities; the patient may

experience intolerable discomfort or pain.

Adverse events will also be graded, by the investigator, for relationship of the AE to study drug. A relationship to study drug category of not related, possible, probable, definite, is defined as

Not Related No temporal association and other etiologies are likely the cause

Possible Temporal association, but other etiologies are likely the cause.

However, involvement of the study drug cannot be excluded.

Probable Temporal association, other etiologies are possible but unlikely. The

event may respond if the study drug is discontinued.

Definite Established temporal association with administration of the study drug

with no other probable cause. The event should resolve when the study

drug is discontinued and recur on re-challenge.

The intensity and relationship assessments to study drug are recorded on the AE CRF page.

Treatment-emergent AEs (TEAEs) will be tabulated, i.e., those events which are not present at baseline or worsened in severity following the start of treatment. Any adverse events starting more than 30 days after the last administration of study drug will not be tabulated.

The onset date of an adverse event will be compared to the date of first dose of study medication in this extension study to determine if the adverse event is treatment emergent

or not. Adverse events with an onset date on or after the date of first dose of study medication will be classified as treatment emergent.

The following adverse event summaries will be provided:

- A summary of the number and percentage of patients reporting a treatment emergent adverse event by body system, and preferred term
- A summary of the number and percentage of patients reporting a treatment emergent adverse event by maximum intensity, body system and preferred term
- A summary of the number and percentage of patients reporting a treatment emergent adverse event by relationship to study drug, body system and preferred term
- A summary of the number and percentage of patients reporting a treatment emergent adverse event leading to dose modification by body system and preferred term

For each patient and each adverse event, the worst severity recorded will be attributed and used in the by-severity summaries. Similarly, the worst causality (most related to treatment) will be attributed and used in the by-causality summaries. If severity or causality are missing, the worst case will be assumed.

The date the AE started should be well collected in CRF data. However, in the unlikely case that the AE start date is missing, the AE date will imputed be as follows.

| | Scenarios | | Imputed AE Onset Date |
|---|---|---|---|
| Day | Month | Year | |
| missing | | | If the month and year of the AE are the same as the month and year of the first dose date in the extension, use the day of the first dose date. |
| | | | Otherwise use 1 for day. |
| | missing | | If year of onset of AE is before the year of first dose in the extension, use DEC. |
| | | | If the year of the AE is the same as the year of the first dose date in the extension and the day of the AE is greater or equal to the day of the first dose in the extension, use the month from the first dose date. If the day of the AE is less than the day of the first dose in the extension, use the month of first dose + 1. If the month of the first dose in the |

Filename: 87272 304 SAP v2 final

| | | | extension is DEC, then use month of first dose. If the year of onset of AE is after the year |
|---|---|---|---|
| | | missing | of first dose in the extension, use JAN. If the day and month of the AE is before the day and month of the first dose in the extension, assign the missing year as the year of the first dose date + 1. Otherwise, assign the missing year as the year of the first dose date. |
| missing | missing | | If year of onset of AE is before the year of first dose in the extension, use 01/07/yyyy. |
| | | | If the year of the AE is the same as the year of the first dose in the extension, use the first dose date. |
| | | | If year of onset of AE is after the year of first dose in the extension, use 01/01/yyyy. |
| | missing | missing | If the day of the AE is before the day of the first dose in the extension, assign the missing month as the month of the first dose date + 1 and the year as the year of the first dose date. If the month of the first dose in the extension is DEC, then +1 year and use JAN. |
| | | | If the day of the AE is on or after the date of the first dose in the extension, assign the missing month and year as the month and year of the first dose date. |
| missing | | missing | If the month of the AE is the same or after<br>the month of the first dose in the<br>extension, then use the day and year from<br>first dose. |
| | | | Otherwise, impute the missing day as 1 |

| | | | and assign the year of the first dose + 1. |
|---------|---------|---------|--------------------------------------------|
| missing | missing | missing | Use the first dose date in the extension. |

A by-patient listing of all adverse events (including non-treatment-emergent events) will be provided. This listing will be presented by treatment group and will include: centre, patient identifier, age, sex, race, adverse event (body system, preferred term, reported term), date of onset, date of resolution, duration, severity, seriousness, action taken, outcome and causality.

# 4.5.3 Deaths, Serious Adverse Events, and Other Significant Adverse Events

A serious adverse event (SAE) is any AE occurring at any dose that results in any of the following outcomes:

- Death
- Is a life-threatening experience. Life-threatening means that the patient was, in the view of the investigator, at immediate risk of death from the event as it occurred
- Requires in-patient hospitalization or prolongation of existing hospitalization. Hospitalization for elective treatment or a pre-existing condition that did not worsen during the clinical investigation is not considered an AE.
- Results in a persistent or significant disability/incapacity (i.e., a substantial disruption of a person's ability to conduct normal life functions). Disability is defined as a substantial disruption in a person's ability to conduct normal life functions
- Results in a congenital anomaly/birth defect

Important medical events that may not result in death, be life threatening, or require hospitalization may be considered SAEs only when they jeopardize the health of the patient or require medical or surgical intervention to prevent one of the outcomes listed in the above definition. If there is any doubt whether the information constitutes an SAE, the information is treated as an SAE in this study.

The following adverse event summaries will be provided:

- A summary of the number and percentage of patients reporting a fatal treatment emergent adverse event by body system, and preferred term
- A summary of the number and percentage of patients reporting a serious treatment emergent adverse event by body system, and preferred term
- A summary of the number and percentage of patients reporting a treatment emergent adverse event leading to withdrawal from the study by body system and preferred term

The following adverse event listings will also be provided:

- A by-patient listing of all deaths that occurred during the study
- A by-patient listing of all serious adverse events
- A by-patient listing of all adverse events leading to withdrawal

#### 4.5.4 Clinical Laboratory Evaluation

All clinical laboratory assessments are implemented by a central laboratory.

The clinical laboratory data were collected at baseline, Months 1, 3, 6, 9, 12, 16, 20, 24, 28, 32, and 36. Additional hematological assessments are collected at Months 2, 4, 8 and 10.

The laboratory data include:

- 1. Hematology: hemoglobin, hematocrit, RBC count, WBC count with differential, and platelet count.
- 2. Blood chemistries: sodium, potassium, chloride, bicarbonate, glucose, cholesterol, creatinine, calcium, phosphorus, BUN, uric acid, total bilirubin, total protein, AST, ALT, and alkaline phosphatase levels.
- 3. Routine urinalysis: specific gravity, pH, protein/albumin, glucose/sugar, ketones/acetone, and hemoglobin/blood. In order to standardize measurements, Bayer multistix 8-SG or equivalent dipsticks will be used.
- 4. Microscopic urinalysis: RBC, WBC, casts, and crystals/cells.

Descriptive statistics for laboratory results and change from baseline for each visit will be presented separately for hematology, biochemistry and urinalysis parameters. The number of patients with clinically significant liver function tests will also be presented.

A by-patient listing of all laboratory data will also be provided with abnormal values highlighted, and including centre, patient identifier, age, sex, race, weight and visit. A listing of the central laboratory reference ranges will also be provided.

# 4.5.5 Vital Signs, Physical Findings and Other Observations Related to Safety

#### 4.5.5.1 Vital Sign Measurements

Vital sign measurements, including supine and standing measurements of systolic blood pressure (mmHg), diastolic blood pressure (mmHg), pulse (bpm), weight (kg), and oral

temperature (°C), are collected at each visit during the open-label extension with the exception of the haematological evaluation visits (Months 2, 4, 8 and 10).

Descriptive statistics for vital sign results and change from baseline for each visit will be presented.

The number of patients with orthostatic hypotension will also be presented. Orthostatic hypotension is defined as either a systolic blood pressure decrease of  $\geq$ 20 mmHg upon standing or a diastolic blood pressure decrease of  $\geq$ 10 mmHg upon standing.

A by-patient listing of all vital sign measurements will also be provided.

#### 4.5.5.2 ECG

The ECG parameters assessment includes heart rate, PR interval, QRS interval, QT interval, and QTc interval.

QT intervals will be corrected using both Bazett's and Fridericia's formulas. For purposes of data analysis, Fridericia's QT correction will be considered as primary. The QT interval and QTc interval data will be presented both as analysis of central tendency (e.g. means, medians) and categorical analyses.

Categorical analysis of QT/QTc interval data are based on the number and percentage of patients meeting or exceeding the limit value that is defined in ICH guideline E14 <sup>[1]</sup>, i.e. Absolute QTc interval prolongation if QTc interval >450, >480, or >500 msec and Change from baseline in QTc interval >30 or >60 msec.

A listing of patients meeting or exceeding the highest limit value, i.e. QTc interval >500 msec or change from baseline in QTc interval >60 msec, will be provided. The listing of patients will include the dose of study medications that the patient was taking on the day prior to the ECG reading.

Descriptive statistics for QT/QTc intervals will be first presented in the tables. The number and percentage of patients for the QT/QTc category in ICH guideline E14 will be presented in the tables, and the patients who have significant QT/QTc measures will be provided in the listings. The means and standard deviations of QT/QTc intervals by week and the patient with significant QT/QTc changes will be also presented in the tables.

A by-patient listing of all ECG data will also be provided.

#### 4.5.5.3 Physical and Neurological Examination

A complete physical examination and complete neurological examination was performed at baseline and at Months 12, 24, and 36. Brief neurological examinations were also performed at all other visits during the open-label extension.

For the 15 items of complete physical exam and 42 items of complete neurological exam, the number and percentage of patients with normal or abnormal results will be presented.

A by-patient listing of physical and neurological examination data will also be provided.

## 4.5.5.4 AUA Symptom Index

An AUA Symptoms Index, a 7-item Likert-scored scale describing urinary bladder function, is completed by the investigator at the baseline phase, and at Months 1, 3 and 12.

Descriptive statistics (n, mean, std, median, minimum, maximum) of the AUA symptom index scores in each treatment group will be presented by two table layouts: 1) AUA raw overall scores at baseline, Months 1, 3 and 12, 2) change from baseline to Month 1, 2 and 12.

Besides the descriptive statistics tables, AUA symptom index scores will be categorized by using 3 levels: 0-7 as mild, 8-19 as moderate, and >19 as severe. A shift table of the number (%) of patients in the categories of mild, moderate, and severe will be provided.

A listing of AUA symptom index data will be provided.

## 4.5.5.5 Post-void Residual (PVR) Bladder Ultrasound

PVR bladder ultrasound data are collected at baseline, and at Months 1, 3 and 12 to assess the patient's bladder function.

Descriptive statistics for the PVR bladder ultrasound results and change from baseline at each visit will be presented. The number and percentage of patients with abnormal PVR bladder ultrasound at each visit will also be presented.

In addition, PVR bladder ultrasound scores will be categorized by using 3 levels: >50ml, >100ml and >150ml will also be provided.

A by-patient listing of the PVR Bladder Ultrasound data will also be provided.

#### 4.5.6 Concomitant Medications

Any on-going medications, including prescription and non-prescription as well as vitamins and herbal supplements, and any new medications taken during the study should be recorded on the Concomitant Medication Record form. The concomitant medications will be coded according to the World Health Organization (WHO) Drug Dictionary. The number and percentage of concomitant medications will be summarized in tables.

A by-patient listing of all concomitant medications will also be provided.

## 4.6 Quality of Life in Epilepsy (QOLIE-31-P)

The patient-weighted 31-item questionnaire (QOLIE-31-P, version 2.0) was administered in this study, describing health-related quality of life in people with epilepsy. The QOLIE-31-P form will be completed by the patient at baseline phase and at Months 3, 6, 9, 12, 24, and 36. Subscale and total scores will be calculated and the subscales grouped into two factors: emotional/psychological effects (seizure worry, overall QOL, emotional well-being, energy/fatigue subscales) and medical/social effects (medication effects, work-driving-social limits, cognitive function subscales).

Descriptive statistics of the QOLIE-31-P data will be presented in the tables and listings for

- Overall assessment
- Emotional/Psychological Effects domain
- Medical/Social Effects domain.

## 4.7 Determination of Sample Size

All participants who have successfully completed the Maintenance and Transition phases of Study VRX-RET-E22-302, for the treatment of partial-onset seizures are eligible (up to approximately 510 patients).

#### 4.8 Changes in the Conduct of the Study or Planned Analysis

No changes in the conduct of the study or planned analysis have occurred.

#### 5 REFERENCES

[1] ICH Steering Committee, "The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-antiarrythmic Drugs, E14", 12 May 2005.

#### **6 REPORTING OUTPUT**

All outputs will be produced using SAS® version 9.1.3 or a later version (if available at PAREXEL). The REPORT procedure will be used to produce all tables and listings whenever possible. The GPLOT procedure will be used to produce all figures whenever possible. All statistical appendices (supportive SAS output) will be output directly from the appropriate SAS procedure.

Valeant Pharmaceuticals North America VRX-RET-E22-304

RM2009/00475/00 VRX-<del>REISTA 221304</del> Plan Version 2.0 [Final]

Post-text tables, listings and statistical appendices will be produced as RTF files using ODS and Courier New font size 9. Figures will be produced as RTF files using ODS and font=simplex. For all outputs, the page numbering will be applied to ensure that when the RTF files are combined, the page numbering remains fixed.

Filename: 87272\_304\_SAP\_v2\_final 

#### 7 LIST OF TABLES

- TABLE 1 NUMBER (%) OF PATIENTS WHO DISCONTINUED TREATMENT DURING THERAPY PHASE BY PRIMARY REASON
- TABLE 2 TIME UNTIL TREATMENT DISCONTINUATION (DAYS)
  DESCRIPTIVE STATISTICS
- TABLE 3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS
- TABLE 4 EPILEPSY HISTORY
- TABLE 5 CLINICAL GLOBAL IMPRESSION (CGI) SEVERITY AT BASELINE
- TABLE 6 NUMBER OF BACKGROUND AEDs AT BASELINE N (%)
- TABLE 7 PRESENCE OF PARTIAL SEIZURE BY SUBTYPE DURING BASELINE PERIOD
- TABLE 9.1 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 1 MONTH DURING THE OPEN-LABEL EXTENSION
- TABLE 9.2 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 3 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.3 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 6 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.4 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 9 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.5 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 12 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.6 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 16 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.7 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 20 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.8 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 24 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.9 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 28 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.10 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 32 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 9.11 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 36 MONTHS DURING THE OPEN-LABEL EXTENSION

- TABLE 10 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY)
- TABLE 11.1 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 1 MONTH DURING THE OPEN-LABEL EXTENSION
- TABLE 11.2 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 3 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.3 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 6 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.4 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 9 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.5 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 12 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.6 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 16 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.7 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 20 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.8 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 24 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.9 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 28 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.10 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 32 MONTHS DURING THE OPEN-LABEL EXTENSION
- TABLE 11.11 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 36 MONTHS DURING THE OPEN-LABEL EXTENSION

- TABLE 12 PROPORTION OF PATIENTS EXPERIENCING A REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY
- TABLE 13 PROPORTION OF SEIZURE-FREE DAYS
- TABLE 14 EXTENT OF EXPOSURE TO STUDY MEDICATION
- TABLE 15 NUMBER (%) OF PATIENTS REPORTING TREATMENT-EMERGENT ADVERSE EVENTS
- TABLE 16 NUMBER (%) OF PATIENTS REPORTING ADVERSE EVENTS BY MAXIMUM SEVERITY
- TABLE 17 NUMBER (%) OF PATIENTS REPORTING TREATMENT-EMERGENT ADVERSE EVENTS AT LEAST POSSIBLY RELATED TO STUDY DRUG
- TABLE 18 NUMBER (%) OF PATIENTS REPORTING TREATMENT-EMERGENT ADVERSE EVENTS THAT LEAD TO DOSE MODIFICATION/INTERRUPTION
- TABLE 19 NUMBER (%) OF PATIENTS REPORTING FATAL TREATMENT-EMERGENT ADVERSE EVENTS
- TABLE 20 NUMBER (%) OF PATIENTS REPORTING SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS
- TABLE 21 NUMBER (%) OF PATIENTS REPORTING ADVERSE EVENTS THAT CAUSED WITHDRAWAL FROM STUDY
- TABLE 22 OBSERVED MEANS AND STANDARD DEVIATIONS OF LABORATORY TEST RESULTS AND CHANGE FROM BASELINE BY MONTH SERUM CHEMISTRY
- TABLE 24 OBSERVED MEANS AND STANDARD DEVIATIONS OF LABORATORY TEST RESULTS AND CHANGE FROM BASELINE BY MONTH HEMATOLOGY
- TABLE 25 OBSERVED MEANS AND STANDARD DEVIATIONS OF LABORATORY TEST RESULTS AND CHANGE FROM BASELINE BY MONTH – URINALYSIS
- TABLE 23 NUMBER (%) OF PATIENTS WITH CLINICALLY SIGNIFICANT LIVER FUNCTION TEST RESULTS
- TABLE 26 FREQUENCY DISTRIBUTION OF CATEGORICAL LABORATORY TEST RESULTS URINALYSIS
- TABLE 27 SUMMARY STATISTICS OF ELECTROCARDIOGRAM MEASURES
- TABLE 28 NUMBER (%) OF PATIENTS EXAMINING QTC INTERVAL BY CATEGORY
- TABLE 29 NUMBER (%) OF PATIENTS EXAMINING QTC INTERVAL CHANGE FROM BASELINE BY CATEGORY
- TABLE 30 OBSERVED MEANS AND STANDARD DEVIATIONS OF QTC INTERVALS AND CHANGE FROM BASELINE BY MONTH
- TABLE 31 OBSERVED MEANS AND STANDARD DEVIATIONS OF VITAL SIGN RESULTS AND CHANGE FROM BASELINE BY MONTH
- TABLE 33 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF PHYSICAL EXAMINATIONS
- TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS
- TABLE 35 NUMBER (%) OF PATIENTS WITH ABNORMAL AUA SYMPTOM INDEX

Valeant Pharmaceuticals North America VRX-RET-E22-304

RM2009/00475/00 VRX-<del>RESTA 221304</del> Plan Version 2.0 [Final]

- TABLE 36 DESCRIPTIVE STATISTICS OF RAW OVERALL AUA SCORES TABLE 37 NUMBER (%) OF PATIENTS WHO HAD MILD, MODERATE, SEVERE
  - **AUA SCORES**
- TABLE 38 AUA CATEGORY SHIFT FROM BASELINE
- TABLE 39 NUMBER (%) OF PATIENTS WITH ABNORMAL PVR BLADDER ULTRASOUND
- TABLE 40 DESCRIPTIVE STATISTICS OF PVR BLADDER ULTRASOUND
- TABLE 41 NUMBER (%) OF PATIENTS WITH A CLINICALLY SIGNIFICANT PVR BLADDER ULTRASOUND
- TABLE 42 NUMBER (%) OF PATIENTS TAKING CONCOMITANT MEDICATIONS
- TABLE 43 OBSERVED MEANS AND STANDARD DEVIATIONS OF QOL IN EPILEPSY (QOLIE-31-P) AND CHANGE FROM BASELINE BY MONTH

Filename: 87272 304 SAP v2 final

# **8 LIST OF FIGURES**

FIGURE 1 MEDIAN PERCENT REDUCTION FROM BASELINE IN SEIZURE FREQUENCY OVER TIME BY DURATION OF TREATMENT EXPOSURE

Filename: 87272\_304\_SAP\_v2\_final 

#### 9 LIST OF PATIENT DATA LISTINGS

- LISTING 1 PATIENT WITHDRAWAL/STUDY COMPLETION
- LISTING 2 INCLUSION/EXCLUSION CRITERIA/ELIGIBILITY
- LISTING 3 DEMOGRAPHICS AND BASELINE CHARACTERISTICS
- LISTING 4 STUDY MEDICATION COMPLIANCE
- LISTING 5 CONCOMITANT MEDICATIONS EXCLUDING BACKGROUND ANTI-EPILEPTIC DRUGS (AEDs)
- LISTING 6 CONCOMITANT TREATMENTS OTHER THAN MEDICATION
- LISTING 7 PARTIAL SEIZURE FREQUENCY
- LISTING 8 GENERALIZED OR UNCLASSIFIED SEIZURE FREQUENCY
- LISTING 9 EXTENT OF EXPOSURE TO STUDY MEDICATION
- LISTING 10 ADVERSE EVENTS CODING DICTIONARY MAPPING
- LISTING 11 ADVERSE EVENTS
- LISTING 12 TREATMENT-EMERGENT ADVERSE EVENTS
- LISTING 13 TREATMENT-EMERGENT ADVERSE EVENTS AT LEAST POSSIBLY RELATED TO STUDY MEDICATION
- LISTING 14 TREATMENT-EMERGENT ADVERSE EVENTS THAT CAUSED WITHDRAWAL FROM STUDY
- LISTING 15 TREATMENT-EMERGENT ADVERSE EVENTS THAT LEAD TO DOSE MODIFICATION/INTERRUPTION
- LISTING 16 DEATHS
- LISTING 17 SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS
- LISTING 18 LABORATORY REFERENCE RANGES
- LISTING 19 HEMATOLOGY LABORATORY TEST RESULTS
- LISTING 20 BLOOD SERUM CHEMISTRY LABORATORY TEST RESULTS
- LISTING 21 URINALYSIS LABORATORY TEST RESULTS
- LISTING 22 ECG DIAGNOSIS/COMMENTS INFORMATION
- LISTING 23 ECG RESULTS
- LISTING 24 ECGS NOT PERFORMED AND THEIR REASON FOR NOT PERFORMING
- LISTING 25 ECG RESULTS FOR PATIENTS WITH QTC INTERVAL >500MSEC OR CHANGE FROM BASELINE IN QTC INTERVAL >60MSEC
- LISTING 26 VITAL SIGNS
- LISTING 27 ABNORMAL PHYSICAL EXAMINATION RESULTS
- LISTING 28 ABNORMAL NEUROLOGICAL EXAMINATION RESULTS
- LISTING 29 AUA SYMPTOM INDEX
- LISTING 30 PVR BLADDER ULTRASOUND RESULTS

Valeant Pharmaceuticals North America VRX-RET-E22-304

RM2009/00475/00 VRX-<del>RESTA 221304</del> Plan Version 2.0 [Final]

LISTING 31 QUALITY OF LIFE IN EPILEPSY SCORES (QOLIE-31-P)

Filename: 87272\_304\_SAP\_v2\_final

RM2009/00475/00 VRX-RET-E22-304

10 TABLE SHELLS

 $\frac{\omega}{2}$ 

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 1 NUMBER (%) OF PATIENTS WHO DISCONTINUED TREATMENT DURING THERAPY PHASE BY PRIMARY REASON SAFETY POPULATION

| | RETIGABINE<br>(N=XXX) |
|---|---|
| DISCONTINUED ANY REASON | xx (xx.x%) |
| ADVERSE EVENT<br>UNSATISFACTORY RESPONSE - EFFICACY | xx (xx.x%)<br>xx (xx.x%) |
| PREGNANT UNWILLING OR UNABLE TO CONTINUE THE STUDY | xx (xx.x%)<br>xx (xx.x%) |
| NON-COMPLIANT WITH STUDY PROCEDURES REQUIRES MEDICATION NOT ALLOWED IN THE PROTOCOL CLINICALLY SIGNIFICANT CHANGE IN MEDICAL CONDITION | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| PERSISTENT ALT OR AST ABOVE 3×ULN ALT OR AST ABOVE 5×ULN AT ANY TIME | xx (xx.x%)<br>xx (xx.x%) |
| CONFIRMED QTC PROLONGATION INVESTIGATOR DECISION | xx (xx.x%)<br>xx (xx.x%) |
| SPONSOR REQUEST FAILURE TO RETURN PATIENT REQUEST UNRELATED TO STUDY | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| OTHER EVENT | xx (xx.x%) |

Program Path/sas program name

32

Run Date:

Filename: 87272\_304\_SAP\_v2\_final

PAGE X OF X

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

# TABLE 2 TIME UNTIL TREATMENT DISCONTINUATION (DAYS) DESCRIPTIVE STATISTICS SAFETY POPULATION

| X |
|----|
| XX |
| X |
| 2 |

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS SAFETY POPULATION

| | RETIGABINE |
|-----------------------------------------|-------------|
| STATISTICS | (N=XXX) |
| AGE - YEAR | |
| N I I I I I I I I I I I I I I I I I I I | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |
| SEX - N (%) | |
| MALE | xxx (xx.x%) |
| FEMALE | xxx (xx.x%) |
| RACE - N (%) | |
| CAUCASIAN | xxx (xx.x%) |
| AFRICAN-AMERICAN (BLACK) | xxx (xx.x%) |
| HISPANIC | xxx (xx.x%) |
| ASIAN | xxx (xx.x%) |
| OTHER | xxx (xx.x%) |
| HEIGHT - CM | |
| N | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |
| WEIGHT - KG | |
| N | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |

Program Path/sas program name

Run Date:

Filename: 87272\_304\_SAP\_v2\_final

PAGE X OF X

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

# TABLE 3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS SAFETY POPULATION

| STATISTICS | RETIGABINE<br>(N=XXX) |
|----------------|-----------------------|
| BMI - (KG/M^2) | |
| N | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |


RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 4 EPILEPSY HISTORY SAFETY POPULATION

| TYPE OF EPILEPSY | RETIGABINE |
|-----------------------------|------------|
| STATISTICS | (N=XXX) |
| PARTIAL (PRIMARY DIAGNOSIS) | |
| DURATION - YEARS | |
| N | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |
| GENERALISED | |
| DURATION - YEARS | |
| N | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |

Program Path/sas program name

36

Run Date:

Filename: 87272\_304\_SAP\_v2\_final


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### FOOTNOTES:

A PATIENT CAN HAVE EPILESPY HISTORY RECORDED FOR EACH TYPE OF EPILEPSY.

3

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Run Date:
Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 5 CLINICAL GLOBAL IMPRESSION (CGI) - SEVERITY AT BASELINE SAFETY POPULATION

| (N=XXX) |
|-------------|
| XXX |
| XXX.X |
| XXX.XX |
| XXX.X |
| XXX |
| XXX |
| xxx (xx.x%) |
| xxx (xx.x%) |
| xxx (xx.x%) |
| xxx (xx.x%) |
| xxx (xx.x%) |
| xxx (xx.x%) |
| xxx (xx.x%) |
| xxx (xx.x%) |

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 6 NUMBER OF BACKGROUND AEDS AT BASELINE N (%) SAFETY POPULATION

| | RETIGABINE |
|------------------------------|-------------|
| CATEGORY | (N=XXX) |
| NUMBER OF AEDs | |
| 1 | xxx (xx.x%) |
| 2 | xxx (xx.x%) |
| 3 | xxx (xx.x%) |
| VAGAL NERVE STIMULATOR USED? | |
| YES | xxx (xx.x%) |
| NO | xxx (xx.x%) |

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 7 PRESENCE OF PARTIAL SEIZURE BY SUBTYPE DURING BASELINE PERIOD SAFETY POPULATION

| CATEGORY | RETIGABINE<br>(N=XXX) |
|------------------------------------------------------|-----------------------|
| BASELINE PERIOD | |
| N | XXX |
| SIMPLE PARTIAL SEIZURES WITH MOTOR SIGNS | xxx (xx.x%) |
| SIMPLE PARTIAL SEIZURES WITHOUT MOTOR SIGNS | xxx (xx.x%) |
| SIMPLE PARTIAL SEIZURES WITH AND WITHOUT MOTOR SIGNS | xxx (xx.x%) |
| COMPLEX PARTIAL SEIZURES | xxx (xx.x%) |
| PARTIAL SEIZURES EVOLVING TO SECONDARY GENERALISED | xxx (xx.x%) |

Program Path/sas program name

40

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

FOOTNOTES: A PATIENT CAN APPEAR IN MULTIPLE CATEGORIES.

4

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 8 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY SAFETY POPULATION

#### RETIGABINE

| | | (N=XXX) | |
|------------------|----------|-------------|-------------------|
| | | CHANGE FROM | PERCENTAGE CHANGE |
| STATISTICS | OBSERVED | BASELINE | FROM BASELINE |
| BASELINE [1] | | | |
| N | xxx | | |
| MEAN | XXX.X | | |
| STD | XXX.XX | | |
| MEDIAN | XXX.X | | |
| MININUM | XXX | | |
| MAXIMUM | xxx | | |
| OPEN-LABEL PHASE | | | |
| N | xxx | xxx | xxx |
| MEAN | XXX.X | XXX.X | xxx.x |
| STD | XXX.XX | XXX.XX | xxx.xx |
| MEDIAN | XXX.X | xxx.x | xxx.x |
| MININUM | XXX | xxx | XXX |
| MAXIMUM | XXX | XXX | XXX |

Program Path/sas program name

42

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

#### FOOTNOTE:

[1] BASELINE PHASE IN STUDY VRX-RET-E22-302

1

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 9.1 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 1 MONTH

DURING THE OPEN-LABEL EXTENSION

SAFETY POPULATION

#### RETIGABINE

| | | (N=XXX) | |
|--------------|----------|-------------|-------------------|
| | | CHANGE FROM | PERCENTAGE CHANGE |
| STATISTICS | OBSERVED | BASELINE | FROM BASELINE |
| BASELINE [1] | | | |
| N | XXX | | |
| MEAN | XXX.X | | |
| STD | XXX.XX | | |
| MEDIAN | XXX.X | | |
| MININUM | XXX | | |
| MAXIMUM | XXX | | |
| MONTH 1 | | | |
| N | XXX | XXX | XXX |
| MEAN | XXX.X | XXX.X | XXX.X |
| STD | XXX.XX | xxx.xx | XXX.XX |
| MEDIAN | XXX.X | xxx.x | xxx.x |
| MININUM | XXX | xxx | XXX |
| MAXIMUM | XXX | XXX | xxx |

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

FOOTNOTE: [1] BASELINE PHASE IN STUDY VRX-RET-E22-302


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name

45

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 9.2 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 3 MONTHS

DURING THE OPEN-LABEL EXTENSION

SAFETY POPULATION

RETIGABINE

| | | (N=XXX) | |
|---|---|---|---|
| | | CHANGE FROM | PERCENTAGE CHANGE |
| STATISTICS | OBSERVED | BASELINE | FROM BASELINE |
| BASELINE [1] | | | |
| N IN | | | |
| MEAN | XXX | | |
| STD | XXX • X | | |
| | XXX.XX | | |
| MEDIAN | XXX.X | | |
| MININUM | XXX | | |
| MAXIMUM | XXX | | |
| MONTH 1 | | | |
| N | xxx | xxx | XXX |
| MEAN | XXX.X | XXX.X | xxx.x |
| STD | XXX.XX | XXX.XX | xxx.xx |
| MEDIAN | xxx.x | xxx.x | xxx.x |
| MININUM | xxx | xxx | xxx |
| MAXIMUM | xxx | XXX | XXX |
| MONTH 3 | | | |
| N | xxx | xxx | xxx |
| MEAN | xxx.x | xxx.x | xxx.x |
| STD | xxx.xx | xxx.xx | xxx.xx |
| MEDIAN | XXX.X | xxx.x | xxx.x |
| MININUM | XXX | XXX | XXX |
| MAXIMUM | XXX | XXX | XXX |

Program Path/sas program name

46

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

FOOTNOTE: [1] BASELINE PHASE IN STUDY VRX-RET-E22-302

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Use Template for TABLE 9.2 to produce:

DURING THE OPEN-LABEL EXTENSION

48

TABLE 9.3 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 6 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.4 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 9 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.5 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 12 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.6 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 16 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.7 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 20 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.8 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 24 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.9 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 28 MONTHS DURING THE OPEN-LABEL EXTENSION TABLE 9.10 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 32 MONTHS DURING THE OPEN-LABEL EXTENSION

PROGRAMMING NOTE: EVERY TIMEPOINT SHOULD BE INCLUDED WITHIN THE INDICATED DURATION OF OPEN-LABEL TREATMENT. E.G. MONTHS 1, 3, 6, 9, 12, 16, 20, 24, 28, 32 AND 36 WILL BE PRESENTED IN TABLE 9.11.

TABLE 9.11 PERCENTAGE CHANGE IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 36 MONTHS

Program Path/sas program name

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 10 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) SAFETY POPULATION

| RESPONSE CATEGORY | RETIGABINE<br>(N=XXX) |
|-----------------------------------|--------------------------------|
| N<br>RESPONDERS<br>NON-RESPONDERS | xx<br>xx (xx.x%)<br>xx (xx.x%) |

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America
Protocol Number: VRX-RET-E22-304

TABLE 11.1 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 1 MONTH DURING THE OPEN-LABEL EXTENSION SAFETY POPULATION

| RESPONSE CATEGORY | RETIGABINE<br>(N=XXX) |
|-------------------|-----------------------|
| MONTH 1 | |
| N | XX |
| RESPONDERS | xx (xx.x%) |
| NON-RESPONDERS | xx (xx.x%) |

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 11.2 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 3 MONTHS DURING THE OPEN-LABEL EXTENSION SAFETY POPULATION

| | RETIGABINE |
|-------------------|------------|
| RESPONSE CATEGORY | (N=XXX) |
| MONTH 1 | |
| N | XX |
| RESPONDERS | xx (xx.x%) |
| NON-RESPONDERS | xx (xx.x%) |
| MONTH 3 | |
| N | XX |
| RESPONDERS | xx (xx.x%) |
| NON-RESPONDERS | xx (xx.x%) |

Program Path/sas program name

57

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

Use Template for TABLE 9.2 to produce:

TABLE 11.3 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT

LEAST 6 MONTHS DURING THE OPEN-LABEL EXTENSION

TABLE 11.4 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 9 MONTHS DURING THE OPEN-LABEL EXTENSION

TABLE 11.5 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT

LEAST 12 MONTHS DURING THE OPEN-LABEL EXTENSION
TABLE 11.6 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT

LEAST 16 MONTHS DURING THE OPEN-LABEL EXTENSION

TABLE 11 7 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SETZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABLINE FOR AT

TABLE 11.7 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 20 MONTHS DURING THE OPEN-LABEL EXTENSION

TABLE 11.8 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 24 MONTHS DURING THE OPEN-LABEL EXTENSION

TABLE 11.9 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT

LEAST 28 MONTHS DURING THE OPEN-LABEL EXTENSION
TABLE 11.10 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT

TABLE 11.10 RESPONDER RATE (>=30% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 32 MONTHS DURING THE OPEN-LABEL EXTENSION

TABLE 11.11 RESPONDER RATE (>=50% REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY) FOR PATIENTS TREATED WITH RETIGABINE FOR AT LEAST 36 MONTHS DURING THE OPEN-LABEL EXTENSION

PROGRAMMING NOTE: EVERY TIMEPOINT SHOULD BE INCLUDED WITHIN THE INDICATED DURATION OF OPEN-LABEL TREATMENT. E.G. MONTHS 1, 3, 6, 9, 12, 16, 20, 24, 28, 32 AND 36 WILL BE PRESENTED IN TABLE 11.11.

Program Path/sas program name

52

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

TABLE 12 PROPORTION OF PATIENTS EXPERIENCING A REDUCTION IN MONTHLY TOTAL PARTIAL SEIZURE FREQUENCY SAFETY POPULATION

| CATEGORY | RETIGABINE<br>(N=XXX) |
|--------------------|-----------------------|
| REDUCTION CATEGORY | |
| [-100%, -75%] | xx (xx.x%) |
| (- 75%, -50%] | xx (xx.x%) |
| (- 50%, -25%] | xx (xx.x%) |
| (- 25%, 0%) | xx (xx.x%) |
| WITHOUT REDUCTION | xx (xx.x%) |

RM2009/00475/00 VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 13 PROPORTION OF SEIZURE-FREE DAYS SAFETY POPULATION

| | RETIGABINE |
|-------------------------------------|------------|
| STATISTICS | (N=XXX) |
| SEIZURE-FREE DAYS (%) | |
| N | XXX |
| MEAN | XXX.X |
| STD | XXX.XX |
| MEDIAN | XXX.X |
| MININUM | XXX |
| MAXIMUM | XXX |
| REDUCTION CATEGORY | |
| SEIZURE-FREE [=100%] | xx (xx.x%) |
| NOT SEIZURE-FREE | xx (xx.x%) |
| [95%, 100%) | xx (xx.x%) |
| [75%, 95%) | xx (xx.x%) |
| [50%, 75%) | xx (xx.x%) |
| [50%, 25%) | xx (xx.x%) |
| [0%, 25%) | xx (xx.x%) |
| NUMBER OF PATIENTS WHO WERE SEIZURE | -FREE FOR |
| 6 MONTHS | xx (xx.x%) |
| 12 MONTHS | xx (xx.x%) |

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 14 EXTENT OF EXPOSURE TO STUDY MEDICATION SAFETY POPULATION

| EXTENT OF EXPOSURE (DAYS) N KEAN MEAN MEAN MEDIAN MININUM MAXIMUM RETIGABINE EXPOSURE CATEGORY (MONTHS) N (1, 3] (3, 6] (4, 9) (5, 9) (12, 16] (12, 16] (12, 16] (14, 20) (15, 20) (16, 20) (20, 24) (20, 24) (20, 24) (24, 28) (24, 28) (24, 28) DAILY DOSE OF RETIGABINE EXPOSURE (MG) N MEAN MEAN MEAN MEAN MININUM MAXIMUM XXX XXX XXX XXX XXX XXX XXX | | RETIGABINE |
|---|---|---|
| N | STATISTICS | (N=XXX) |
| N | | |
| MEAN XXX.XX STD XXX.XX MEDIAN XXX MININUM XXX MAXIMUM XXX RETIGABINE EXPOSURE CATEGORY (MONTHS) XXX (100.0%) [0, 1] XXX (XX.X%) (1, 3] XXX (XX.X%) (3, 6] XXX (XX.X%) (6, 9] XXX (XX.X%) (12, 16] XXX (XX.X%) (12, 16] XXX (XX.X%) (20, 24] XXX (XX.X%) (24, 28] XXX (XX.X%) (24, 28] XXX (XX.X%) (32, 36] XXX (XX.X%) >36 XXX DAILY DOSE OF RETIGABINE EXPOSURE (MG) XXX N XXX MEAN XXX.X MEDIAN XXX.X MININUM XXX | , , | |
| STD | | |
| MEDIAN | | |
| MININUM | | |
| MAXIMUM xxx RETIGABINE EXPOSURE CATEGORY (MONTHS) N xxx (100.0%) [0, 1] xxx (xx.x%) (1, 3] xxx (xx.x%) (3, 6] xxx (xx.x%) (6, 9] xxx (xx.x%) (9, 12] xxx (xx.x%) (12,16] xxx (xx.x%) (16,20] xxx (xx.x%) (20,24] xxx (xx.x%) (24,28] xxx (xx.x%) (28,32] xxx (xx.x%) (32,36] xxx (xx.x%) >36 xxx DAILY DOSE OF RETIGABINE EXPOSURE (MG) xxx N xxx MEAN xxx.x STD xxx.xx MEDIAN xxx.x MININUM xxx | | |
| RETIGABINE EXPOSURE CATEGORY (MONTHS) N | | |
| N | MAXIMUM | XXX |
| N | RETIGABINE EXPOSURE CATEGORY (MONTHS) | |
| [0, 1] | | xxx (100.0%) |
| (1, 3] | [0, 1] | |
| (3, 6] | | |
| (6, 9] | | |
| (9, 12] | | |
| (12,16] xxx (xx.x%) (16,20] xxx (xx.x%) (20,24] xxx (xx.x%) (24,28] xxx (xx.x%) (28,32] xxx (xx.x%) (32,36] xxx (xx.x%) >36 xxx DAILY DOSE OF RETIGABINE EXPOSURE (MG) xxx N xxx MEAN xxx.x STD xxx.xx MEDIAN xxx.xx MININUM xxx | | XXX ( XX.X%) |
| (16,20] | | XXX ( XX.X%) |
| (20,24] xxx (xx.x%) (24,28] xxx (xx.x%) (28,32] xxx (xx.x%) (32,36] xxx (xx.x%) >36 xxx (xx.x%) DAILY DOSE OF RETIGABINE EXPOSURE (MG) xxx N xxx MEAN xxx.x STD xxx.xx MEDIAN xxx.xx MININUM xxx.x | | XXX ( XX.X%) |
| (24,28] xxx (xx.x%) (28,32] xxx (xx.x%) (32,36] xxx (xx.x%) >36 xxx (xx.x%) DAILY DOSE OF RETIGABINE EXPOSURE (MG) xxx N xxx MEAN xxx.x STD xxx.xx MEDIAN xxx.x MININUM xxx | | xxx ( xx.x%) |
| (32,36] | (24,28] | XXX ( XX.X%) |
| (32,36] | (28, 32] | XXX ( XX.X%) |
| DAILY DOSE OF RETIGABINE EXPOSURE (MG) N | | XXX ( XX.X%) |
| N xxx MEAN xxx.x STD xxx.xx MEDIAN xxx.x MININUM xxx | >36 | |
| N xxx MEAN xxx.x STD xxx.xx MEDIAN xxx.x MININUM xxx | DATLY DOSE OF PETTCABINE EXPOSIDE (MC) | |
| MEAN xxx.x STD xxx.xx MEDIAN xxx.x MININUM xxx | , , | XXX |
| STD | | |
| MEDIAN XXX.X<br>MININUM XXX | | |
| MININUM xxx | | |
| | MAXIMUM | XXX |

Program Path/sas program name

55

Run Date:

CONFIDENTIAL RM

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### TABLE 15 NUMBER (%) OF PATIENTS REPORTING TREATMENT-EMERGENT ADVERSE EVENTS SAFETY POPULATION

| SYSTEM ORGAN CLASS | RETIGABINE |
|------------------------|--------------|
| PREFERRED TERM | (N=XXX) |
| ANY ADVERSE EVENT | xxx ( xx.x%) |
| 1ST SYSTEM ORGAN CLASS | xxx ( %x.x%) |
| PREFERRED TERMS BELOW | xxx ( xx.x%) |
| 2ND SYSTEM ORGAN CLASS | xxx ( xx.x%) |
| PREFERRED TERMS BELOW | xxx ( xx.x%) |

Program Path/sas program name

56

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 16 NUMBER (%) OF PATIENTS REPORTING ADVERSE EVENTS BY MAXIMUM SEVERITY SAFETY POPULATION

| SYSTEM ORGAN CLASS | | | |
|------------------------|----------------------|--------------|--------------|
| PREFERRED TERM | MILD | MODERATE | SEVERE |
| 1ST SYSTEM ORGAN CLASS | (8x.xx ) xxx (8x.xx) | xxx ( xx.x%) | xxx ( xx.x%) |
| PREFERRED TERMS BELOW | | xxx ( xx.x%) | xxx ( xx.x%) |
| 2ND SYSTEM ORGAN CLASS | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| PREFERRED TERMS BELOW | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

Program Path/sas program name

Run Date:


RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

col Number: VRX-RET-E22-304

Use Template for TABLE 15 to produce:

TABLE 17 NUMBER (%) OF PATIENTS REPORTING TREATMENT-EMERGENT ADVERSE EVENTS AT LEAST POSSIBLY RELATED TO STUDY DRUG TABLE 18 NUMBER (%) OF PATIENTS REPORTING TREATMENT-EMERGENT ADVERSE EVENTS THAT LEAD TO DOSE MODIFICATION/INTERRUPTION

TABLE 19 NUMBER (%) OF PATIENTS REPORTING FATAL TREATMENT-EMERGENT ADVERSE EVENTS

TABLE 20 NUMBER (%) OF PATIENTS REPORTING SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS

TABLE 21 NUMBER (%) OF PATIENTS REPORTING ADVERSE EVENTS THAT CAUSED WITHDRAWAL FROM STUDY

Program Path/sas program name

Ö.

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 22 OBSERVED MEANS AND STANDARD DEVIATIONS OF LABORATORY TEST RESULTS AND CHANGE FROM BASELINE BY MONTH - SERUM CHEMISTRY SAFETY POPULATION

| | | RETIGABINE<br>(N=XXX) | | |
|---|---|---|---|---|
| | | | | Change from |
| | | | | Baseline |
| TEST NAME (TEST UNIT) | TIMEPOINT | n | Mean (STD) | Mean (STD) |
| | _ | | | |
| SODIUM (MMOL/L) | BASELINE | XXX | xx.x (xx.xx) | |
| | MONTH 1 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 16 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 20 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 28 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 32 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 36 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| POTASSIUM (MMOL/L) | : | | | |

Use Template for TABLE 22 to produce:

TABLE 24 OBSERVED MEANS AND STANDARD DEVIATIONS OF LABORATORY TEST RESULTS AND CHANGE FROM BASELINE BY MONTH - HEMATOLOGY TABLE 25 OBSERVED MEANS AND STANDARD DEVIATIONS OF LABORATORY TEST RESULTS AND CHANGE FROM BASELINE BY MONTH - URINALYSIS

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

#### TABLE 23 NUMBER (%) OF PATIENTS WITH CLINICALLY SIGNIFICANT LIVER FUNCTION TEST RESULTS SAFETY POPULATION

| UNIT) | TIMEPOINT | n | >3xULN | >5xULN | >10xULN |
|--------------|-----------|-----|--------------|--------------|-------------|
| ALT (MMOL/L) | BASELINE | xxx | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 1 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 16 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 20 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 28 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 32 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | MONTH 36 | XXX | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |

REPEAT FOR TOTAL BILIRUBIN AND ALKALINE PHOSPHATASE

Program Path/sas program name

Run Date:


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 26 FREQUENCY DISTRIBUTION OF CATEGORICAL LABORATORY TEST RESULTS - URINALYSIS SAFETY POPULATION

| RETI | GABINE |
|------|--------|
| /37 | |

| | (N=XXX) | |
|-----------|-----------------------------------------|----------|
| | | <u> </u> |
| TEST NAME | | |
| MONTH 1 | | |
| 1+ | xx (xx.x%) | |
| 2+ | xx (xx.x%) | |
| 3+ | xx (xx.x%) | |
| 4+ | xx (xx.x%) | |
| - ' | *************************************** | |
| MONTH 3 | | |
| 1+ | xx (xx.x%) | |
| 2+ | xx (xx.x%) | |
| 3+ | xx (xx.x%) | |
| 4+ | xx (xx.x%) | |
| | , , , , | |
| MONTH 6 | | |
| MONTH 9 | | |
| MONTH 12 | | |
| MONTH 16 | | |
| MONTH 20 | | |
| MONTH 24 | | |
| MONTH 28 | | |
| MONTH 32 | | |
| MONTH 36 | | |

REPEAT FOR ALL NON-NUMERIC TEST RESULTS

Program Path/sas program name

<u>ი</u>

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### TABLE 27 SUMMARY STATISTICS OF ELECTROCARDIOGRAM MEASURES SAFETY POPULATION

| | EVALUATION - UNIT | RETIGABINE |
|--------------|----------------------------|------------|
| TIMEPOINT | STATISTIC | (N=XXX) |
| BASELINE AVG | VENTRICULAR RATE - BPM | |
| DASELINE AVG | N N VENTRICULAR RAIL - BPM | |
| | MEAN | XXX |
| | MEAN<br>STD | XXX.X |
| | | XXX.XX |
| | MEDIAN | XXX.X |
| | MINIMUM | XXX |
| | MAXIMUM | XXX |
| | RR INTERVAL - MS | |
| | N | XXX |
| | MEAN | XXX.X |
| | STD | xxx.xx |
| | MEDIAN | xxx.x |
| | MINIMUM | XXX |
| | MAXIMUM | xxx |
| | PR INTERVAL - MS | |
| | N | XXX |
| | MEAN | XXX.X |
| | STD | XXX.XX |
| | MEDIAN | XXX.X |
| | MINIMUM | XXX |
| | MAXIMUM | xxx |
| | ORS INTERVAL - MS | |
| | N N | xxx |
| | MEAN | XXX.X |
| | STD | XXX.XX |
| | MEDIAN | |
| | MEDIAN<br>MINIMUM | XXX.X |
| | | XXX |
| | MAXIMUM | XXX |

Program Path/sas program name

62

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 27 SUMMARY STATISTICS OF ELECTROCARDIOGRAM MEASURES SAFETY POPULATION

| TIMEPOINT | EVALUATION - UNIT<br>STATISTIC | RETIGABINE<br>(N=XXX) |
|---|---|---|
| BASELINE AVG (CONTINUED) | OT INTERVAL - MS | |
| Discipling MVG (CONTINODD) | N PIO | XXX |
| | MEAN | XXX.X |
| | STD | XXX.XX |
| | MEDIAN | XXX.X |
| | MINIMUM | XXX |
| | MAXIMUM | |
| | MAXIMUM | XXX |
| | OTC INTERVAL BAZETT - MS | |
| | N<br>N | XXX |
| | MEAN | xxx.x |
| | STD | xxx.xx |
| | MEDIAN | xxx.x |
| | MINIMUM | XXX |
| | MAXIMUM | xxx |
| | OTC INTERVAL FRIDERICIA - MS | |
| | N | xxx |
| | MEAN | XXX.X |
| | STD | XXX.XX |
| | MEDIAN | XXX.X |
| | MINIMUM | |
| | MINIMUM<br>MAXIMUM | xxx |

REPEAT FOR TIMEPOINTS MONTH 1, MONTH 3, MONTH 6, MONTH 9, MONTH 12, MONTH 24, MONTH 36

Program Path/sas program name

63

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 28 NUMBER (%) OF PATIENTS EXAMINING QTC INTERVAL BY CATEGORY SAFETY POPULATION

| TIMEPOINT | CATEGORY | RETIGABINE<br>(N=XXX) |
|---|---|---|
| BASELINE AVG (CONTINUED) | ABSOLUTE QTc INTERVAL (MS) | |
| | FRIDERICIA'S CORRECTION | |
| | <= 450 | xx (xx.x%) |
| | (450, 480] | xx (xx.x%) |
| | (480, 500] | xx (xx.x%) |
| | > 500 | xx (xx.x%) |
| | BAZETT'S CORRECTION | |
| | <= 450 | xx (xx.x%) |
| | (450, 480] | xx (xx.x%) |
| | (480, 500] | xx (xx.x%) |
| | > 500 | xx (xx.x%) |

REPEAT FOR TIMEPOINTS MONTH 1, MONTH 3, MONTH 6, MONTH 9, MONTH 12, MONTH 24, MONTH 36

Program Path/sas program name

64

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 29 NUMBER (%) OF PATIENTS EXAMINING QTC INTERVAL CHANGE FROM BASELINE BY CATEGORY SAFETY POPULATION

| TIMEPOINT | CATEGORY | RETIGABINE<br>(N=XXX) |
|---|---|---|
| MONTH 1 | CHANGE FROM BASELINE IN QTc INTERVAL (MS) FRIDERICIA'S CORRECTION <= 30 (30, 60] > 60 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| | BAZETT'S CORRECTION <= 30 (30, 60] > 60 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

REPEAT FOR TIMEPOINTS MONTH 3, MONTH 6, MONTH 9, MONTH 12, MONTH 24, MONTH 36

Program Path/sas program name

65

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 30 OBSERVED MEANS AND STANDARD DEVIATIONS OF QTC INTERVALS AND CHANGE FROM BASELINE BY MONTH SAFETY POPULATION

| | RETIGABINE<br>(N=XXX) | | |
|---|---|---|---|
| TIMEPOINT | n | Mean (STD) | Change from<br>Baseline<br>Mean (STD) |
| ABSOLUTE QTc (FRIDERICIA'S) INTERVAL (MS) | | | |
| MONTH 1 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 36 | xxx | xx.x (xx.xx) | xx.x (xx.xx) |
| ABSOLUTE QTc (BAZETT'S) INTERVAL (MS) | | | |
| MONTH 1 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MONTH 36 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |

Program Path/sas program name

66

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 31 OBSERVED MEANS AND STANDARD DEVIATIONS OF VITAL SIGN RESULTS AND CHANGE FROM BASELINE BY MONTH SAFETY POPULATION

| | | | RETIGABINE<br>(N=XXX) | |
|---|---|---|---|---|
| | <del></del> | | <u>`</u> | |
| PARAMETER (PARAMETER UNIT) | TIMEPOINT | n | Mean (STD) | Mean (STD) |
| SUPINE SBP (MMHG) | BASELINE | xxx | xx.x (xx.xx) | |
| | MONTH 1 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 16 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 20 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 28 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 32 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 36 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| SUPINE DBP (MMHG) | : | | | |

Program Path/sas program name

Run Date:

0

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 32 NUMBER (%) OF PATIENTS WITH ORTHOSTATIC HYPOTENSION SAFETY POPULATION

| TIMEPOINT | | RETIGABINE<br>(N=XXX) |
|-----------|-----|-----------------------|
| BASELINE | N | xx |
| | YES | xx (xx.x%) |
| | NO | xx (xx.x%) |
| MONTH 1 | N | xx |
| | YES | xx (xx.x%) |
| | NO | xx (xx.x%) |
| MONTH 3 | N | xx |
| | YES | xx (xx.x%) |
| | NO | xx (xx.x%) |
| MONTH 6 | N | xx |
| | YES | xx (xx.x%) |
| | NO | xx (xx.x%) |
| MONTH 9 | N | xx |
| | YES | xx (xx.x%) |
| | NO | xx (xx.x%) |
| MONTH 12 | N | xx |
| | YES | xx (xx.x%) |
| | NO | xx (xx.x%) |

REPEAT FOR TIMEPOINTS MONTH 16, MONTH 20, MONTH 24, MONTH 28, MONTH 32 AND MONTH 36

#### FOOTNOTES:

ORTHOSTATIC HYPOTENSION IS DEFINED AS EITHER A DECREASE IN SBP>=20 MMHG UPON STANDING OR DECREASE IN DBP>=10 MMHG UPON STANDING

Program Path/sas program name Run Date:

Valeant Pharmaceuticals North America

Protocol Number: VRX-RET-E22-304

PAGE X OF X

Ç

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# Table 33 Number (%) of patients with abnormal results of physical examinations safety population

| TIMEPOINT | PHYSICAL<br>EXAMINATION | | RETIGABINE<br>(N=XXX) |
|---|---|---|---|
| BASELINE | SKIN | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | HEAD | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | EYES | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | EARS | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | NOSE | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | THROAT | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | MOUTH | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | NECK | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | CHEST | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | HEART | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | | | \ <i>-</i> , |

REPEAT FOR TIMEPOINTS MONTH 12, MONTH 24 AND MONTH 36

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### TABLE 33 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF PHYSICAL EXAMINATIONS SAFETY POPULATION

| TIMEPOINT | PHYSICAL<br>EXAMINATION | | RETIGABINE<br>(N=XXX) |
|---|---|---|---|
| BASELINE | LUNGS | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | BREAST | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | ABDOMEN | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | GENITALIA | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | EXTREMITIES | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | OTHER | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |

REPEAT FOR TIMEPOINTS MONTH 12, MONTH 24 AND MONTH 36

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS SAFETY POPULATION

| TIMEPOINT | | | RETIGABINE<br>(N=XXX) |
|---|---|---|---|
| BASELINE | NEUROLOGICAL EXAMINATION - COMPLETE<br>GENERAL | | |
| | LEVEL OF CONSCIOUSNESS | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | LEVEL OF APPEARANCE/MOTOR EXPRESSION | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | MENTAL STATUS | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | SPEECH | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | CRANIAL NERVES<br>VISION | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | EYE MOVEMENTS | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | JAW MOVEMENT AND FACIAL SENSATION | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | FACIAL MOTOR | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | SWALLOWING, PHARYNX, LARYNX | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | STERNOCLEIDOMASTOID, TRAPEZIUS | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |
| | TONGUE | NORMAL<br>ABNORMAL | xx (xx.x%)<br>xx (xx.x%) |

Program Path/sas program name

72

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS SAFETY POPULATION

| AL XX ( AL XX ( AL XX ( XX ( XX ( XX ( | xx.x%)<br>xx.x%)<br>xx.x%)<br>xx.x%)<br>xx.x%)<br>xx.x%)<br>xx.x%) |
|---|---|
| AL XX ( AL XX ( AL XX ( XX ( XX ( XX ( | xx.x%) xx.x%) xx.x%) xx.x%) xx.x%) |
| XX ( AL XX ( AL XX ( XX ( | xx.x%) xx.x%) xx.x%) xx.x%) xx.x%) |
| AL XX ( AL XX ( XX ( | xx.x%) xx.x%) xx.x%) xx.x%) |
| xx ( | xx.x%)<br>xx.x%)<br>xx.x%) |
| AL xx ( | xx.x%)<br>xx.x%) |
| xx ( | xx.x%) |
| , | * |
| AL XX ( | xx.x%) |
| xx ( | xx.x%) |
| AL xx ( | xx.x%) |
| xx ( | xx.x%) |
| AL xx ( | xx.x%) |
| xx ( | xx.x%) |
| AL xx ( | xx.x%) |
| xx ( | xx.x%) |
| AL XX ( | xx.x%) |
| | xx.x%) |
| AL xx ( | xx.x%) |
| | xx.x%) |
| xx ( | xx.x%) |
| | xx ( |

Program Path/sas program name

Run Date:
Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS SAFETY POPULATION

| | | | RETIGABINE |
|---|---|---|---|
| TIMEPOINT | | | (N=XXX) |
| BASELINE | NEUROLOGICAL EXAMINATION - COMPLETE MUSCLE STRENGTH | | |
| | TRUNK | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | UPPER EXTREMITIES | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | LOWER EXTREMITIES | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | MUSCLE TONE | | |
| | UPPER EXTREMITIES | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | LOWER EXTREMITIES | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | COORDINATION/CEREBELLAR FUNCTION | | |
| | GAIT | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | HOPPING | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | ROMBERG | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | NYSTAGMUS | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | TREMOR | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS SAFETY POPULATION

| TIMEPOINT | | | RETIGABINE<br>(N=XXX) |
|---|---|---|---|
| BASELINE | NEUROLOGICAL EXAMINATION - COMPLETE COORDINATION/CEREBELLAR FUNCTION | | |
| | FINGER-NOSE | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | HEEL-SHIN | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | RAPID RHYTHMIC MOVEMENTS | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | SENSATION: UPPER EXTREMITIES | | |
| | PAIN/TEMPERATURE | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | LIGHT TOUCH | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | POSITION | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | VIBRATION | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | SENSATION: LOWER EXTREMITIES | | |
| | PAIN/TEMPERATURE | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | LIGHT TOUCH | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |

Program Path/sas program name

75

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS SAFETY POPULATION

| TIMEPOINT | | | RETIGABINE<br>(N=XXX) |
|---|---|---|---|
| BASELINE | NEUROLOGICAL EXAMINATION - COMPLETE<br>SENSATION: LOWER EXTREMITIES | | |
| | POSITION | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | VIBRATION | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| MONTH 1 | NEUROLOGICAL EXAMINATION - BRIEF GENERAL | | |
| | LEVEL OF CONSCIOUSNESS | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | MENTAL STATUS | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | REFLEXES | | |
| | BICEPS | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | KNEE | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | MOTOR SYSTEM | | |
| | GENERAL MOVEMENT | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |

Program Path/sas program name

76

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### TABLE 34 NUMBER (%) OF PATIENTS WITH ABNORMAL RESULTS OF NEUROLOGICAL EXAMINATIONS SAFETY POPULATION

| TIMEPOINT | | | RETIGABINE<br>(N=XXX) |
|---|---|---|---|
| MONTH 1 | NEUROLOGICAL EXAMINATION - BRIEF COORDINATION/CEREBELLAR FUNCTION | | |
| | GAIT | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | HOPPING | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | ROMBERG | NORMAL | xx (xx.x%) |
| | ROIBERG | ABNORMAL | xx (xx.x%) |
| | NYSTAGMUS | NORMAT | xx (xx.x%) |
| | NISIAGMOS | ABNORMAL | xx (xx.x%) |
| | | | ( |
| | TREMOR | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | FINGER-NOSE | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | HEEL-SHIN | NORMAL | xx (xx.x%) |
| | | ABNORMAL | xx (xx.x%) |
| | RAPID RHYTHMIC MOVEMENTS | NORMAL | xx (xx.x%) |
| | | | . , |

REPEAT IN ORDER OF VISITS USING THE PROPER FORMAT OF COMPLETE OR BRIEF DEPENDING UPON VISIT IE. BASELINE (COMPLETE), MONTH 1 (BRIEF), MONTH 3 (BRIEF), MONTH 6 (BRIEF), MONTH 9 (BRIEF), MONTH 12 (COMPLETE), MONTH 16 (BRIEF), MONTH 20 (BRIEF), MONTH 24 (COMPLETE), MOTH 28 (BRIEF), MONTH 32 (BRIEF), MONTH 36 (COMPLETE)

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## TABLE 35 NUMBER (%) OF PATIENTS WITH ABNORMAL AUA SYMPTOM INDEX SAFETY POPULATION

| | | RETIGABINE |
|---|---|---|
| CIMEPOINT | | (N=XXX) |
| BASELINE | 1. HOW OFTEN HAVE YOU HAD A SENSATION OF NOT EMPTYING YOUR BLADDER COMPLETELY? | |
| 110221112 | NOT AT ALL | xx (xx.x%) |
| | LESS THAN 1 TIME IN 5 | xx (xx.x%) |
| | LESS THAN HALF TIME | xx (xx.x%) |
| | ABOUT HALF THE TIME | xx (xx.x%) |
| | MORE THAN HALF THE TIME | xx (xx.x%) |
| | ALMOST ALWAYS | xx (xx.x%) |
| | 2. HOW OFTEN HAVE YOU HAS TO URINATE AGAIN LESS THAN 2 HOURS AFTER YOU FINISHED URINATING? | |
| | NOT AT ALL | xx (xx.x%) |
| | LESS THAN 1 TIME IN 5 | xx (xx.x%) |
| | LESS THAN HALF TIME | xx (xx.x%) |
| | ABOUT HALF THE TIME | xx (xx.x%) |
| | MORE THAN HALF THE TIME | xx (xx.x%) |
| | ALMOST ALWAYS | xx (xx.x%) |
| | 3. HOW OFTEN HAVE YOU FOUND YOU STOPPED AND STARTED AGAIN SEVERAL TIMES WHEN YOU URINATED? | |
| | NOT AT ALL | xx (xx.x%) |
| | LESS THAN 1 TIME IN 5 | xx (xx.x%) |
| | LESS THAN HALF TIME | xx (xx.x%) |
| | ABOUT HALF THE TIME | xx (xx.x%) |
| | MORE THAN HALF THE TIME | xx (xx.x%) |
| | ALMOST ALWAYS | xx (xx.x%) |
| | 4. HOW OFTEN HAVE YOU FOUND IT DIFFICULT TO POSTPONE URINATION? | |
| | NOT AT ALL | xx (xx.x%) |
| | LESS THAN 1 TIME IN 5 | xx (xx.x%) |
| | LESS THAN HALF TIME | xx (xx.x%) |
| | ABOUT HALF THE TIME | xx (xx.x%) |
| | MORE THAN HALF THE TIME | xx (xx.x%) |
| | ALMOST ALWAYS | xx (xx.x%) |

Program Path/sas program name

78

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## TABLE 35 NUMBER (%) OF PATIENTS WITH ABNORMAL AUA SYMPTOM INDEX SAFETY POPULATION

| TIMEPOINT | | RETIGABINE<br>(N=XXX) |
|---|---|---|
| BASELINE | 5. HOW OFTEN HAVE YOU HAD A WEAK URINARY STREAM? | |
| | NOT AT ALL | xx (xx.x%) |
| | LESS THAN 1 TIME IN 5 | xx (xx.x%) |
| | LESS THAN HALF TIME | xx (xx.x%) |
| | ABOUT HALF THE TIME | xx (xx.x%) |
| | MORE THAN HALF THE TIME | xx (xx.x%) |
| | ALMOST ALWAYS | xx (xx.x%) |
| | 6. HOW OFTEN HAVE YOU HAD TO PUSH OR STRAIN TO BEGIN URINATION? | |
| | NOT AT ALL | xx (xx.x%) |
| | LESS THAN 1 TIME IN 5 | xx (xx.x%) |
| | LESS THAN HALF TIME | xx (xx.x%) |
| | ABOUT HALF THE TIME | xx (xx.x%) |
| | MORE THAN HALF THE TIME | xx (xx.x%) |
| | ALMOST ALWAYS | xx (xx.x%) |
| | 7. HOW MANY TIMES DID YOU MOST TYPICALLY GET UP TO URINATE FROM THE TIME YOU WENT TO BED UNTIL THE TIME YOU GOT UP? | |
| | NONE | xx (xx.x%) |
| | 1 TIME | xx (xx.x%) |
| | 2 TIMES | xx (xx.x%) |
| | 3 TIMES | xx (xx.x%) |
| | 4 TIMES | xx (xx.x%) |
| | 5 TIMES OR MORE | xx (xx.x%) |
| | | (/ |

REPEAT FOR TIMEPOINTS MONTH 1, MONTH 3 AND MONTH 12

Program Path/sas program name

Run Date:

80

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

## TABLE 36 DESCRIPTIVE STATISTICS OF RAW OVERALL AUA SCORES SAFETY POPULATION

#### RETIGABINE

| | | (N=XXX) | |
|-------------|------------|----------|-------------|
| | | OBSERVED | CHANGE FROM |
| TIMEPOINT | STATISTICS | | BASELINE |
| BASELINE | N | XXX | |
| 21102221112 | MEAN | xxx.x | |
| | STD | xxx.xx | |
| | MEDIAN | XXX.X | |
| | MINIMUM | XXX | |
| | MAXIMUM | XXX | |
| MONIBII 1 | N | | |
| MONTH 1 | N | XXX | XXX |
| | MEAN | XXX.X | XXX.X |
| | STD | XXX.XX | XXX.XX |
| | MEDIAN | XXX.X | XXX.X |
| | MINIMUM | XXX | XXX |
| | MAXIMUM | XXX | XXX |
| MONTH 3 | N | XXX | XXX |
| | MEAN | XXX.X | XXX.X |
| | STD | XXX.XX | XXX.XX |
| | MEDIAN | XXX.X | XXX.X |
| | MINIMUM | xxx | xxx |
| | MAXIMUM | XXX | XXX |
| MONTH 12 | N | XXX | XXX |
| | MEAN | xxx.x | XXX.X |
| | STD | xxx.xx | XXX.XX |
| | MEDIAN | xxx.x | XXX.X |
| | MINIMUM | xxx | XXX |
| | MAXIMUM | xxx | xxx |

Program Path/sas program name

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 37 NUMBER (%) OF PATIENTS WHO HAD MILD, MODERATE, SEVERE AUA SCORES SAFETY POPULATION

| TIMEPOINT | CATEGORY | RETIGABINE<br>(N=XXX) |
|---|---|---|
| BASELINE | N<br>MILD [0,7]<br>MODERATE [8,19]<br>SEVERE (>19) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 1 | N<br>MILD [0,7]<br>MODERATE [8,19]<br>SEVERE (>19) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 3 | N<br>MILD [0,7]<br>MODERATE [8,19]<br>SEVERE (>19) | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 3 | N<br>MILD [0,7]<br>MODERATE [8,19]<br>SEVERE (>19) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

Program Path/sas program name

 $\infty$ 

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

#### TABLE 38 AUA CATEGORY SHIFT FROM BASELINE SAFETY POPULATION

#### RETIGABINE

| | | (N=XXX) | |
|-----------------|------------|----------------|--------------|
| FROM BASELINE | MILD [0,7] | MODERATE[8,19] | SEVERE (>19) |
| TO MONTH 1 | | | |
| TO MONTH 1 | | | |
| MILD [0,7] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MODERATE [8,19] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SEVERE (>19) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TO MONTH 3 | | | |
| MILD [0,7] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MODERATE [8,19] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SEVERE (>19) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| TO MONTH 12 | | | |
| MILD [0,7] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MODERATE [8,19] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SEVERE (>19) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | | _ |

Program Path/sas program name

82

Run Date:


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

TABLE 39 NUMBER (%) OF PATIENTS WITH ABNORMAL PVR BLADDER ULTRASOUND SAFETY POPULATION

| TIMEPOINT | CATEGORY | RETIGABINE<br>(N=XXX) |
|-----------|-------------------------|--------------------------------|
| BASELINE | N<br>ABNORMAL<br>NORMAL | xx<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 1 | N<br>ABNORMAL<br>NORMAL | xx<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 3 | N<br>ABNORMAL<br>NORMAL | xx<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 12 | N<br>ABNORMAL<br>NORMAL | xx<br>xx (xx.x%)<br>xx (xx.x%) |

Run Date:


RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## TABLE 40 DESCRIPTIVE STATISTICS OF PVR BLADDER ULTRASOUND SAFETY POPULATION

#### RETIGABINE

| | | (N=XXX) | 1.01101.01 |
|-----------|-----------|---------|----------------------|
| TIMEPOINT | STATISTIC | ACTUAL | CHANGE FROM BASELINE |
| BASELINE | N | xxx | |
| | MEAN | XXX.X | |
| | STD | XXX.XX | |
| | MEDIAN | XXX.X | |
| | MINIMUM | XXX | |
| | MAXIMUM | xxx | |
| MONTH 1 | N | xxx | xxx |
| | MEAN | xxx.x | XXX.X |
| | STD | XXX.XX | XXX.XX |
| | MEDIAN | XXX.X | XXX.X |
| | MINIMUM | xxx | XXX |
| | MAXIMUM | xxx | xxx |
| MONTH 3 | N | xxx | xxx |
| | MEAN | XXX.X | XXX.X |
| | STD | XXX.XX | XXX.XX |
| | MEDIAN | XXX.X | XXX.X |
| | MINIMUM | XXX | XXX |
| | MAXIMUM | xxx | xxx |
| MONTH 12 | N | xxx | xxx |
| | MEAN | XXX.X | XXX.X |
| | STD | xxx.xx | xxx.xx |
| | MEDIAN | XXX.X | XXX.X |
| | MINIMUM | xxx | xxx |
| | MAXIMUM | xxx | xxx |

Program Path/sas program name Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 41 NUMBER (%) OF PATIENTS WITH A CLINICALLY SIGNIFICANT PVR BLADDER ULTRASOUND SAFETY POPULATION

| TIMEPOINT | CATEGORY | RETIGABINE<br>(N=XXX) |
|---|---|---|
| BASELINE | N<br>>50mL<br>>100mL<br>>150mL | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 1 | N<br>>50mL<br>>100mL<br>>150mL | xx<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 3 | N<br>>50mL<br>>100mL<br>>150mL | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| MONTH 12 | N<br>>50mL<br>>100mL<br>>150mL | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

Program Path/sas program name

85

Run Date:

CONFIDENTIAL RM2

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

# TABLE 42 NUMBER (%) OF PATIENTS TAKING CONCOMITANT MEDICATIONS SAFETY POPULATION

| MEDICATION 1 | PREFERRED TE | ERM | | <del></del> | TIGABINE<br>N=XXX) |
|---|---|---|---|---|---|
| CONCOMITANT | MEDICATION | PREFERRED | TERM | XX | (xx.x%) |

Program Path/sas program name

86

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

TABLE 43 OBSERVED MEANS AND STANDARD DEVIATIONS OF QOL IN EPILEPSY (QOLIE-31-P) AND CHANGE FROM BASELINE BY MONTH SAFETY POPULATION

RETIGABINE (N=XXX)

| | | (14-3737 | / | |
|---|---|---|---|---|
| | | | | Change from<br>Baseline |
| CATEGORY | TIMEPOINT | n | Mean (STD) | Mean (STD) |
| OVER 1. 1. O O TO O VEN TO | D. 607 TVD | | , | |
| OVERALL ASSESSMENT | BASELINE | XXX | xx.x (xx.xx) | , |
| | MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 36 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| EMOTIONAL/PYSCHOLOGICAL EFFECTS DOMAIN | BASELINE | xxx | xx.x (xx.xx) | |
| | MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 6 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 9 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 12 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 24 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 36 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| MEDICAL/SOCIAL EFFECTS DOMAIN | BASELINE | xxx | xx.x (xx.xx) | |
| | MONTH 3 | XXX | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 6 | xxx | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 9 | xxx | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 12 | xxx | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 24 | xxx | xx.x (xx.xx) | xx.x (xx.xx) |
| | MONTH 36 | xxx | xx.x (xx.xx) | xx.x (xx.xx) |

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304

11 FIGURE SHELLS

88

FIGURE 1 MEDIAN PERCENT REDUCTION FROM BASELINE IN SEIZURE FREQUENCY OVER TIME BY DURATION OF TREATMENT EXPOSURE SAFETY POPULATION



89

RM2009/00475/00 VRX-RET-E22-304

12 PATIENT DATA LISTING SHELLS

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 1 PATIENT WITHDRAWAL/STUDY COMPLETION

PATIENT ID

INITIALS AGE GENDER RACE

STATUS

DATE OF TAPERING DOSE DISCONTINUED

IF DISCONTINUED,

OR USED?

PRIMARY REASON OF STUDY DRUG DISPENSED DISCONTINUATION

SECONDARY REASON(S) OF DISCONTINUATION

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

#### LISTING 2 INCLUSION/EXCLUSION CRITERIA/ELIGIBILITY

| | | INCLUS | SION C | RITERI | A | EXC | CLUSION C | RITERIA | ELIG | BIBLE |
|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT ID AGE/GENDER/RACE | Q1 | Q2 | Q3 | Q4 | 05 | Q1 | Q2 | Q3 | Q1 | Q2 |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 3 DEMOGRAPHICS AND BASELINE CHARACTERISTICS

| | | | | START DATE | HEIGHT | | CLINICAL | DURATION | TREATMENT/ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | CONSENT | BASELINE | OF EXTENSION | (cm)/ | | GLOBAL | 0F | STUDY | NUMBER OF | |
| PATIENT | | DATE | DATE | STUDY MED. | WEIGHT | BMI | IMPRESSIONS | ILLNESS | DURATION | BACKGROUND | COMPLETED |
| ID | AGE/GENDER/RACE | (STUDY DAY) | (DAY 0) | (STUDY DAY) | (kg) | (kg/m²) | SEVERITY | (YEARS) | (DAYS) | AEDS | STUDY? |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name

96

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### LISTING 4 STUDY MEDICATION COMPLIANCE

| | | | | | | 50 MG | | 100 MG | | 300 MG | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | DATE | DATE | | NUMBER OF | NUMBER | NUMBER OF | NUMBER | NUMBER OF | NUMBER |
| | | | OF | OF | PRESCRIBED | TABLETS | 0F | TABLETS | OF | TABLETS | 0F |
| PATIENT | | | FIRST | LAST | DOSE | DISPENSED | TABLETS | DISPENSED | TABLETS | DISPENSED | TABLETS |
| ID | AGE/GENDER/RACE | STUDY VISIT | DOSE | DOSE | (MG/DAY) | | RETURNED | | RETURNED | | RETURNED |
| This s | ection contained c | lata from each in | dividual | patient, | rather than in | n aggregate. | They have | e been exclu | ided to pro | otect patient | privacy. |
| | nized data from ea | | | | | | | | | | |
| Allollyll | inzed data irom ec | | | | | | | | i fulfiller if | normation p | icase see |
| | | the Pati | ent Leve | Data se | ection of the | Sponsor Cilr | ncai Study | Register. | | | |

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

۶

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 5 CONCOMITANT MEDICATIONS EXCLUDING BACKGROUND ANTI-EPILEPTIC DRUGS (AEDs)

TOTAL DAILY DOSE

PATIENT ID AGE/GENDER/RACE REPORTED TERM PREFERRED TERM PRIMARY ATC CLASSIFICATION AND UNITS START DATE STOP DATE ONGOING?

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

NOTE THIS IS FROM DERIVED CM DATA SET WHERE CMTYPE = 2 AND THE CMREAS is not B or F

NOTE THAT THERE APPEARS TO BE SOME ANTI-EPILEPTIC DRUGS THAT HAVE A CMREAS OTHER THAN B OR F IN THIS LISTING THIS IS BEING MEDICALLY REVIEWED.

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 6 CONCOMITANT TREATMENTS OTHER THAN MEDICATION

PATIENT ID AGE/GENDER/RACE REPORTED TERM

REASON FOR TREATMENT SPECIFY START DATE

STOP DATE ONGOING?

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

NOTE THIS IS FROM DERIVED CT DATA SET WHERE CTTERM IS NOT MISSING

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America

PAGE X OF X

102

Protocol Number: VRX-RET-E22-304

\_\_\_\_

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 7 PARTIAL SEIZURE FREQUENCY

----SIMPLE PARTIAL SEIZURES----

| | | | | | | | | | PARTIAL |
|---|---|---|---|---|---|---|---|---|---|
| | | | DID SEIZURES | | WITH | | COMPLEX | | EVOLVING TO |
| PATIENT | ī | | OCCUR SINCE | DATE OF SEIZURE | MOTOR | WITHOUT MOTOR | PARTIAL | | SECONDARILY |
| ID | AGE/GENDER/RACE | VISIT | LAST VISIT | (STUDY DAY) | SIGNS | SIGNS | SEIZURES | FLURRIES | GENERALIZED |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name

104

Filename: 87272\_304\_SAP\_v2\_final


RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 8 GENERALIZED OR UNCLASSIFIED SEIZURE FREQUENCY

DATE OF

SEIZURE TONIC-PARITAL DID SEIZURES CONVULSIVE PATIENT OCCUR SINCE (STUDY ABSENCE MYOCLONIC CLONIC STATUS STATUS UNCLASSIFIED ID AGE/GENDER/RACE SEIZURES SEIZURES ATONIC EPILEPTICUS **EPILEPTICUS** SEIZURES VISIT LAST VISIT DAY) SEIZURES

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

105

Run Date:

Filename: 87272 304 SAP v2 final

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name

106

107

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### LISTING 9 EXTENT OF EXPOSURE TO STUDY MEDICATION

| | | | | | | AVERAGE DAILY | |
|---|---|---|---|---|---|---|---|
| | | | TREATMENT START | TREATMENT | | DOSE OF STUDY | EXTENT OF |
| PATIENT | | STUDY VISIT | DATE | STOP DATE | TOTAL DOSE (MG) | MEDICATION | EXPOSURE |
| ID | AGE/GENDER/RACE | | | | | (MG/DAY) | (DAYS) |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### LISTING 10 ADVERSE EVENTS CODING DICTIONARY MAPPING

| SYSTEM ORGAN CLASS | PREFERRED TERM | REPORTED TERM |
|--------------------|------------------|-----------------|
| SOC 1 | PREFERRED TERM 1 | REPORTED TERM 1 |
| | | REPORTED TERM 2 |
| | PREFERRED TERM 2 | REPORTED TERM 1 |
| | : | |
| SOC 2 | PREFERRED TERM 1 | REPORTED TERM 1 |
| | | REPORTED TERM 2 |
| | PREFERRED TERM 2 | REPORTED TERM 1 |

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304

Program Path/sas program name
OUTCOME

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

SAE?

LISTING 11 ADVERSE EVENTS

START

DATE

PATIENT REPORTED PREFERRED (STUDY ACTION(S) SITE ID AGE/GENDER/RACE TERM TERM DAY) STOP DATE INTENSITY RELATIONSHIP TAKEN

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

THE FORMAT ABOVE SHOULD BE REPEATED FOR THE FOLLOWING LISTINGS:

LISTING 12 TREATMENT-EMERGENT ADVERSE EVENTS

LISTING 13 TREATMENT-EMERGENT ADVERSE EVENTS AT LEAST POSSIBLY RELATED TO STUDY MEDICATION

LISTING 14 TREATMENT-EMERGENT ADVERSE EVENTS THAT CAUSED WITHDRAWAL FROM STUDY

LISTING 15 TREATMENT-EMERGENT ADVERSE EVENTS THAT LEAD TO DOSE MODIFICATION/INTERRUPTION

LISTING 16 DEATHS

NOTE THAT THIS IS WHERE AEOUT = 4 FATAL IF NO DEATHS THEN 'NONE REPORTED' SHOULD BE DISPLAYED

LISTING 17 SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS

IF NO SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS THEN 'NONE REPORTED' SHOULD BE DISPLAYED

Program Path/sas program name

Run Date:

Filename: 87272 304 SAP v2 final

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Program Path/sas program name

Filename: 87272\_304\_SAP\_v2\_final

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 18 LABORATORY REFERENCE RANGES

NORMAL RANGE NORMAL RANGE
LABORATORY
PARAMETER SI LAB UNIT (SI) (SI)

112

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

-

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

RM20


14

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 19 HEMATOLOGY LABORATORY TEST RESULTS

PLATELET PATIENT COLLECTION DATE WBC RBC HGB HCT LYMPH, ABS COUNT LYMPH ID AGE/GENDER/RACE VISIT (STUDY DAY) X10E3/UL X10E6/UL g/dL % X10E3/UL X10E3/UL

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy.

Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## FOOTNOTES:

\* INDICATES A REPEAT VISIT.

H = HIGH. L = LOW.

Program Path/sas program name

Run Date:


RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 19 HEMATOLOGY LABORATORY TEST RESULTS

| | | | | | MONO, | | EOS, | | BASO, | | NEUI, | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | | | COLLECTION DATE | MONO | ABS, | EOS | ABS | BAS0 | ABS | NEUT | ABS | |
| ID | AGE/GENDER/RACE | VISIT | (STUDY DAY) | % | X10E3/UL | % | X10E3/UL | % | X10E3/UL | % | X10E3/UL | MORPHOLOGY |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## FOOTNOTES:

\* INDICATES A REPEAT VISIT.

H = HIGH. L = LOW.

Program Path/sas program name


RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 20 BLOOD SERUM CHEMISTRY LABORATORY TEST RESULTS

| | | | | ALI | AST | ALK. | 101. | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | | | COLLECTION DATE | SGPT | SGOT | PHOS. | BILI. | CREA. | BUN | CHOL. | PHOS. |
| ID | AGE/GENDER/RACE | VISIT | (STUDY DAY) | IU/L | IU/L | IU/L | mg/dL | mg/dL | md/dL | mg/dL | mg/dL |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy.

Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

Run Date:

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## FOOTNOTES:

\* INDICATES A REPEAT VISIT.

H = HIGH. L = LOW.

Program Path/sas program name


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 20 BLOOD SERUM CHEMISTRY LABORATORY TEST RESULTS

TOT.

PATIENT COLLECTION DATE **GLUCOSE** PROT. URIC ACID Κ Cl BICARBONATE ID AGE/GENDER/RACE VISIT (STUDY DAY) mg/dLg/dL mg/dL mg/dL mEq/L mEq/L mEq/L mEq/L

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

7

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

## FOOTNOTES:

\* INDICATES A REPEAT VISIT.

H = HIGH. L = LOW.

121

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name Run Date:

CONFIDENTIAL RM2

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 21 URINALYSIS LABORATORY TEST RESULTS

**PATIENT** COLLECTION DATE SPEC. WBC RBC LEUK. EPI. AGE/GENDER/RACE VISIT (STUDY DAY) рΗ GRAV. PROTEIN KETONES GLUCOSE BLOOD /HPF /HPF ESTER. BACTERIA CELLS

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Note: This listing should also contain any urinalysis results for crystals.

Program Path/sas program name

122

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

# FOOTNOTES:

\* INDICATES A REPEAT VISIT.

H = HIGH. L = LOW.

123

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name Run Date: 124

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 22 ECG DIAGNOSIS/COMMENTS INFORMATION

PATIENT ID INITIALS AGE/GENDER/RACE VISIT DAY) TIME QUALITY DIAGNOSIS INTERPRETATION ECG COMMENTS

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

the Sponsor Clinical Study Register.

Program Path/sas program name

Run Date:

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

125

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 23 ECG RESULTS

PATIENT ID INITIALS AGE/GENDER/RACE VISIT ECG DATE ECG TIME HR RR PR QRS QT AXIS QTCB QTCF

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

NOTE ONLY RECORDS WITH AT LEAST 1 NON-MISSING RESULT WILL BE PRESENTED IN THIS LISTING

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

12/

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

#### FOOTNOTES:

1 PATIENT HAD AN INTERVAL >500MSEC OR CHANGE FROM BASELINE IN QTC INTERVAL >60MSEC

Program Path/sas program name


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 24 ECGS NOT PERFORMED AND THEIR REASON FOR NOT PERFORMING

PATIENT ID

INITIALS

AGE/GENDER/RACE

VISIT

REASON FOR NOT PERFORMING ECG

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

NOTE ONLY RECORDS WHERE THE VALUE OF THE ECGRES VARIABLE IS NON-MISSING SHOULD BE LISTED HERE.

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

129

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PATIENT ID INITIALS AGE/GENDER/RACE VISIT

LISTING 25 ECG RESULTS FOR PATIENTS WITH QTC INTERVAL >500MSEC OR CHANGE FROM BASELINE IN QTC INTERVAL >60MSEC

TREATMENT DOSE

(MG/DAY)

BEFORE

ECG DATE

**ECG** TIME

ECG

DAY OF ECG

QRS

AXIS

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

NOTE ONLY RECORDS WITH AT LEAST 1 NON-MISSING RESULT WILL BE PRESENTED IN THIS LISTING

RM2009/00475/00 VRX-RET-E22-304


131

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

## FOOTNOTES:

1 PATIENT HAD AN INTERVAL >500MSEC OR CHANGE FROM BASELINE IN QTC INTERVAL >60MSEC

Program Path/sas program name

OTANDINO


3.2

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 26 VITAL SIGNS

| | | | DATE OF VITAL | SUPTINE | SUPTINE | SUPTINE | STANDING | STANDING | STANDING | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | | | SIGNS | SYSTOLIC | DIASTOLIC | PULSE | SYSTOLIC | DIASTOLIC | PULSE | WEIGHT | TEMP. |
| ID | AGE/GENDER/RACE | VISIT | (STUDY DAY) | mmHg | mmHg | bpm | mmHg | mmHg | bpm | kg | °C |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

### FOOTNOTE:

\* INDICATES A >=7% INCREASE IN BODY WEIGHT FROM BASELINE

Ç

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 27 ABNORMAL PHYSICAL EXAMINATION RESULTS

PATIENT DATE OF EXAM

ID AGE/GENDER/RACE VISIT (STUDY DAY) BODY SYSTEM REPORTED ABNORMALITY

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

NOTE UNDER BODY SYSTEM IS THE VALUES OF EITHER THE NON-MISSING PEBODSYS VARIABLE VALUE OR THE PEOTHER VARIABLE VALUE IF PEBODSYS IS MISSING.

RM2009/00475/00 VRX-RET-E22-304


RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Program Path/sas program name

Filename: 87272\_304\_SAP\_v2\_final


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 28 ABNORMAL NEUROLOGICAL EXAMINATION RESULTS

PATIENT ID

AGE/GENDER/RACE VISIT

DATE OF EXAM (STUDY DAY)

EXAM GROUP

GROUP PARAMETER

REPORTED ABNORMALITY

CLINICALLY SIGNIFICANT?

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America

Protocol Number: VRX-RET-E22-304

PAGE X OF X

9

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 29 AUA SYMPTOM INDEX

DATE OF EXAM

PATIENT ID AGE/GENDER/RACE VISIT (STUDY DAY) Q1 Q2 Q3 Q4 Q5 Q6 Q7

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

FOOTNOTES:

QUESTION 1 HOW OFTEN HAVE YOU HAD A SENSATION OF NOT EMPTYING YOUR BLADDER COMPLETELY AFTER YOU FINISHED URINATING?

Program Path/sas program name

Run Date:

8

RM2009/00475/00 VRX-RET-E22-304


S

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

QUESTION 2 HOW OFTEN HAVE YOU HAD TO URINATE AGAIN LESS THAN 2 HOURS AFTER YOU FINISHED URINATING?

QUESTION 3 HOW OFTEN HAVE YOU FOUND YOU STOPPED AND STARTED AGAIN SEVERAL TIMES WHEN YOU URINATED?

QUESTION 4 HOW OFTEN HAVE YOU FOUND IT DIFFICULT TO POSTPONE URINATION?

QUESTION 5 HOW OFTEN HAVE YOU HAD A WEAK URINARY STREAM?

QUESTION 6 HOW OFTEN HAVE YOU HAD TO PUSH OR STRAIN TO BEGIN URINATION?

QUESTION 7 HOW MANY TIMES DID YOU MOST TYPICALLY GET UP TO URINATE FROM THE TIME YOU WENT TO BED AT NIGHT UNTIL THE TIME YOU GOT UP?

Program Path/sas program name

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 30 PVR BLADDER ULTRASOUND RESULTS

DATE OF EXAM

PVR URINE VOLUME

PATIENT ID

AGE/GENDER/RACE

VISIT

(STUDY DAY)

INTERPRETATION

(mL)

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name

14

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Program Path/sas program name

Filename: 87272\_304\_SAP\_v2\_final


142

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 31 QUALITY OF LIFE IN EPILEPSY SCORES (QOLIE-31-P)

PATIENT DATE OF EXAM

ID AGE/GENDER/RACE VISIT (STUDY DAY) Q1 Q2 Q3 Q4 Q5 Q6 Q7 Q8 Q9 Q10 Q11 Q12 Q13 Q14 Q15 Q16 Q17 Q18

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

Run Date:

143

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Program Path/sas program name

Filename: 87272\_304\_SAP\_v2\_final


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 31 QUALITY OF LIFE IN EPILEPSY SCORES (QOLIE-31-P)

| | | | | | PART DPART E | | | | | | | PART F | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PATIENT | | | DATE OF EXAM | | | | | | | | | | | | | | | | | |
| ID | AGE/GENDER/RACE | VISIT | (STUDY DAY) | Q19 | Q20 | Q21 | 022 | Q23 | Q24 | Q25 | Q26 | Q27 | Q28 | Q29 | Q30 | Q31 | Q32 | Q33 | Q34 | Q35 |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name Run Date:

Valeant Pharmaceuticals North America

Protocol Number: VRX-RET-E22-304

PAGE X OF X

145

RM2009/00475/00 VRX-RET-E22-304


Program Path/sas program name


146

RM2009/00475/00 VRX-RET-E22-304

Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

LISTING 31 QUALITY OF LIFE IN EPILEPSY SCORES (QOLIE-31-P)

| | | | | PART G | | PART H | | | | PART I- | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| · | | | DATE OF EXAM | | | | | | | | | | |
| PATIENT ID | AGE/GENDER/RACE | VISIT | (STUDY DAY) | Q36 | Q37 | Q38 | Q39A | Q39B | Q39C | Q39D | Q39E | Q39F | Q39G |

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

14/

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Program Path/sas program name

Filename: 87272\_304\_SAP\_v2\_final


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

LISTING 31 QUALITY OF LIFE IN EPILEPSY SCORES (QOLIE-31-P)

| | | | | | SCORING | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | SEIZURE | | | | | ENERGY | | SOCIAL | | |
| PATIENT | | | DATE OF EXAM | WORRY | OVERALL | EMOTIONAL | FATIGUE | COGNITIVE | MEDICATION | FUNCTIONING | OVERALL |
| ID | AGE/GENDER/RACE | VISIT | (STUDY DAY) | SCORE | QOL SCORE | WELL BEING | SCORE | SCORE | EFFECTS SCORE | SCORE | SCORE |

COORTNO

This section contained data from each individual patient, rather than in aggregate. They have been excluded to protect patient privacy. Anonymized data from each patient may be made available subject to an approved research proposal. For further information please see the Patient Level Data section of the Sponsor Clinical Study Register.

Program Path/sas program name

148

Run Date:

RM2009/00475/00 VRX-RET-E22-304


Valeant Pharmaceuticals North America Protocol Number: VRX-RET-E22-304

PAGE X OF X

Program Path/sas program name

Filename: 87272\_304\_SAP\_v2\_final

